CLINICAL TRIAL: NCT01663402
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Effect of Alirocumab (SAR236553/REGN727) on the Occurrence of Cardiovascular Events in Patients Who Have Recently Experienced an Acute Coronary Syndrome
Brief Title: ODYSSEY Outcomes: Evaluation of Cardiovascular Outcomes After an Acute Coronary Syndrome During Treatment With Alirocumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC11570; 2011-005698-21 (EudraCT Number); U1111-1127-4323 (Other: UTN)
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for alirocumab) subcutaneous (SC) injection every 2 weeks (Q2W) added to stable Lipid-Modifying Therapy (LMT) for up to 64 months.
  Interventions: Drug: Placebo; Drug: LMT
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Experimental): Alirocumab 75 mg SC injection Q2W added to stable LMT for up to 64 months. Alirocumab dose up-titrated to 150 mg Q2W from Month 2 when Low-Density Lipoprotein Cholesterol (LDL-C) levels >=50 mg/dL (1.29 mmol/L) at Month 1; or if up-titration was missed due to unavailability of LDL-C value, it was up-titrated at month 4 based on LDL-C value at Month 2. For participants receiving 150 mg Q2W, alirocumab dose was down-titrated in a blinded manner to 75 mg Q2W if two consecutive values of LDL-C were <25 mg/dL (0.65 mmol/L). For participants receiving 75 mg Q2W, alirocumab dose was switched to placebo in a blinded manner if two consecutive values of LDL-C were <15 mg/dL (0.39 mmol/L).
  Interventions: Drug: Alirocumab; Drug: LMT

INTERVENTIONS:
Drug: Alirocumab — Alirocumab administered as SC injection of 1 mL in the abdomen or thigh with a disposable auto-injector.
  Other Names: SAR236553; REGN727; Praluent®
  Arms: Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Drug: Placebo — Placebo matched to alirocumab administered as a SC injection of 1 mL in the abdomen or thigh with a disposable auto-injector.
  Arms: Placebo
Drug: LMT — Statins (atorvastatin or rosuvastatin) at stable maximal tolerated dose of statin with or without other LMT as clinically indicated.

SUMMARY:
Primary Objective:

To compare the effect of alirocumab with placebo on the occurrence of cardiovascular (CV) events (composite endpoint of coronary heart disease (CHD) death, non-fatal myocardial infarction (MI), fatal and non-fatal ischemic stroke, unstable angina (UA) requiring hospitalization) in participants who experienced an acute coronary syndrome (ACS) event 4 to 52 weeks prior to randomization and were treated with evidence-based medical and dietary management of dyslipidemia.

Secondary Objectives:

* To evaluate the effect of alirocumab on secondary endpoints (any CHD event , major CHD event, any CV event, composite of all cause mortality/non-fatal MI/non-fatal ischemic stroke, CHD deaths, CV deaths, all cause mortality).
* To evaluate the safety and tolerability of alirocumab.
* To evaluate the effect of alirocumab on lipid parameters.

DETAILED DESCRIPTION:
18924 number of participants aged >= 40 years old were randomized in the study.

ELIGIBILITY:
Inclusion criteria :

Recently (< 52 weeks) hospitalized for ACS.

Exclusion criteria:

* Age < 40 years.
* ACS event occurring more than 52 weeks prior to randomization visit.
* LDL-C likely to be <70 mg/dL (<1.81 mmo/L), and apolipoprotein B (ApoB) <80 mg/dL (<0.8 g/L), and non - high-density lipoprotein cholesterol (HDL-C) <100 mg/dL (<2.59 mmol/L) with evidence-based medical and dietary management of dyslipidemia.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18924 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1388):
- United States (273):
  - Investigational Site Number 840163, Birmingham, Alabama
  - Investigational Site Number 840060, Birmingham, Alabama
  - Investigational Site Number 840117, Huntsville, Alabama
  - Investigational Site Number 840192, Huntsville, Alabama
  - Investigational Site Number 840121, Mobile, Alabama
  - Investigational Site Number 840319, Mobile, Alabama
  - Investigational Site Number 840332, Atlantis, Arizona
  - Investigational Site Number 840320, Newport Beach, Arizona
  - Investigational Site Number 840103, Tucson, Arizona
  - Investigational Site Number 840084, Tucson, Arizona
  - Investigational Site Number 840139, Banning, California
  - Investigational Site Number 840286, Beverly Hills, California
  - Investigational Site Number 840246, Beverly Hills, California
  - Investigational Site Number 840353, Beverly Hills, California
  - Investigational Site Number 840341, Carmichael, California
  - Investigational Site Number 840299, Chula Vista, California
  - Investigational Site Number 840164, Fresno, California
  - Investigational Site Number 840076, Fullerton, California
  - Investigational Site Number 840073, Huntington Beach, California
  - Investigational Site Number 840092, La Jolla, California
  - Investigational Site Number 840208, Long Beach, California
  - Investigational Site Number 840068, Long Beach, California
  - Investigational Site Number 840269, Los Alamitos, California
  - Investigational Site Number 840009, Los Angeles, California
  - Investigational Site Number 840282, Los Angeles, California
  - Investigational Site Number 840019, Mission Viejo, California
  - Investigational Site Number 840336, Moreno Valley, California
  - Investigational Site Number 840124, Northridge, California
  - Investigational Site Number 840251, Pasadena, California
  - Investigational Site Number 840289, Pasadena, California
  - Investigational Site Number 840312, Port Hueneme, California
  - Investigational Site Number 840261, San Diego, California
  - Investigational Site Number 840310, San Diego, California
  - Investigational Site Number 840024, San Diego, California
  - Investigational Site Number 840071, Santa Ana, California
  - Investigational Site Number 840236, Santa Rosa, California
  - Investigational Site Number 840012, Torrance, California
  - Investigational Site Number 840096, Aurora, Colorado
  - Investigational Site Number 840037, Colorado Springs, Colorado
  - Investigational Site Number 840189, Denver, Colorado
  - Investigational Site Number 840122, Bridgeport, Connecticut
  - Investigational Site Number 840219, Guilford, Connecticut
  - Investigational Site Number 840347, Altamonte Springs, Florida
  - Investigational Site Number 840066, Clearwater, Florida
  - Investigational Site Number 840079, Daytona Beach, Florida
  - Investigational Site Number 840051, Daytona Beach, Florida
  - Investigational Site Number 840368, Delray Beach, Florida
  - Investigational Site Number 840242, Fort Lauderdale, Florida
  - Investigational Site Number 840134, Gainesville, Florida
  - Investigational Site Number 840327, Hollywood, Florida
  - Investigational Site Number 840153, Hudson, Florida
  - Investigational Site Number 840105, Hudson, Florida
  - Investigational Site Number 840253, Jacksonville, Florida
  - Investigational Site Number 840141, Jacksonville, Florida
  - Investigational Site Number 840042, Jacksonville, Florida
  - Investigational Site Number 840206, Jacksonville, Florida
  - Investigational Site Number 840063, Jacksonville, Florida
  - Investigational Site Number 840002, Jupiter, Florida
  - Investigational Site Number 840119, Largo, Florida
  - Investigational Site Number 840241, Miami Beach, Florida
  - Investigational Site Number 840210, Mount Clemens, Florida
  - Investigational Site Number 840366, New Port Richey, Florida
  - Investigational Site Number 840311, Palm Beach Gardens, Florida
  - Investigational Site Number 840280, Palm Harbor, Florida
  - Investigational Site Number 840054, Panama City, Florida
  - Investigational Site Number 840239, Pembroke Pines, Florida
  - Investigational Site Number 840044, Pensacola, Florida
  - Investigational Site Number 840367, Plantation, Florida
  - Investigational Site Number 840132, Safety Harbor, Florida
  - Investigational Site Number 840061, Safety Harbor, Florida
  - Investigational Site Number 840247, Sarasota, Florida
  - Investigational Site Number 840264, Tampa, Florida
  - Investigational Site Number 840082, Tampa, Florida
  - Investigational Site Number 840213, Trinity, Florida
  - Investigational Site Number 840165, Wellington, Florida
  - Investigational Site Number 840323, West Palm Beach, Florida
  - Investigational Site Number 840075, Atlanta, Georgia
  - Investigational Site Number 840176, Augusta, Georgia
  - Investigational Site Number 840048, Covington, Georgia
  - Investigational Site Number 840065, Cumming, Georgia
  - Investigational Site Number 840356, Thomasville, Georgia
  - Investigational Site Number 840114, Tucker, Georgia
  - Investigational Site Number 840211, Idaho Falls, Idaho
  - Investigational Site Number 840237, Arlington Heights, Illinois
  - Investigational Site Number 840292, Chicago, Illinois
  - Investigational Site Number 840146, Harvey, Illinois
  - Investigational Site Number 840340, Joliet, Illinois
  - Investigational Site Number 840196, Peoria, Illinois
  - Investigational Site Number 840081, Rock Island, Illinois
  - Investigational Site Number 840090, Rock Island, Illinois
  - Investigational Site Number 840358, Elkhart, Indiana
  - Investigational Site Number 840036, Hammond, Indiana
  - Investigational Site Number 840026, Indianapolis, Indiana
  - Investigational Site Number 840102, Muncie, Indiana
  - Investigational Site Number 840145, South Bend, Indiana
  - Investigational Site Number 840154, Ames, Iowa
  - Investigational Site Number 840345, Iowa City, Iowa
  - Investigational Site Number 840283, West Des Moines, Iowa
  - Investigational Site Number 840335, Kansas City, Kansas
  - Investigational Site Number 840089, Kansas City, Kansas
  - Investigational Site Number 840218, Kansas City, Kansas
  - Investigational Site Number 840140, Overland Park, Kansas
  - Investigational Site Number 840030, Lexington, Kentucky
  - Investigational Site Number 840023, Louisville, Kentucky
  - Investigational Site Number 840007, Louisville, Kentucky
  - Investigational Site Number 840279, Owensboro, Kentucky
  - Investigational Site Number 840308, Pikeville, Kentucky
  - Investigational Site Number 840181, Saint Paul, Kentucky
  - Investigational Site Number 840254, Alexandria, Louisiana
  - Investigational Site Number 840344, Lafayette, Louisiana
  - Investigational Site Number 840187, Lake Charles, Louisiana
  - Investigational Site Number 840291, Minden, Louisiana
  - Investigational Site Number 840278, New Orleans, Louisiana
  - Investigational Site Number 840290, Shreveport, Louisiana
  - Investigational Site Number 840142, Auburn, Maine
  - Investigational Site Number 840148, Auburn, Maine
  - Investigational Site Number 840097, Bangor, Maine
  - Investigational Site Number 840234, Framingham, Maine
  - Investigational Site Number 840276, Scarborough, Maine
  - Investigational Site Number 840351, Annapolis, Maryland
  - Investigational Site Number 840072, Beltsville, Maryland
  - Investigational Site Number 840193, Bethesda, Maryland
  - Investigational Site Number 840200, Columbia, Maryland
  - Investigational Site Number 840349, Rockville, Maryland
  - Investigational Site Number 840111, Winfield, Maryland
  - Investigational Site Number 840056, Boston, Massachusetts
  - Investigational Site Number 840144, Flint, Michigan
  - Investigational Site Number 840365, Grandville, Michigan
  - Investigational Site Number 840093, Kalamazoo, Michigan
  - Investigational Site Number 840198, Lansing, Michigan
  - Investigational Site Number 840087, Rochester Hills, Michigan
  - Investigational Site Number 840004, Springfield, Michigan
  - Investigational Site Number 840267, Springfield, Michigan
  - Investigational Site Number 840035, Ypsilanti, Michigan
  - Investigational Site Number 840199, Duluth, Minnesota
  - Investigational Site Number 840116, Edina, Minnesota
  - Investigational Site Number 840281, Minneapolis, Minnesota
  - Investigational Site Number 840094, Saint Cloud, Minnesota
  - Investigational Site Number 840324, Saint Paul, Minnesota
  - Investigational Site Number 840046, Columbia, Missouri
  - Investigational Site Number 840180, Independence, Missouri
  - Investigational Site Number 840013, Marquette, Missouri
  - Investigational Site Number 840179, Overland, Missouri
  - Investigational Site Number 840228, St Louis, Missouri
  - Investigational Site Number 840233, St Louis, Missouri
  - Investigational Site Number 840235, St Louis, Missouri
  - Investigational Site Number 840175, St Louis, Missouri
  - Investigational Site Number 840125, St Louis, Missouri
  - Investigational Site Number 840168, St Louis, Missouri
  - Investigational Site Number 840274, Thomure, Missouri
  - Investigational Site Number 840032, Kalispell, Montana
  - Investigational Site Number 840033, Grand Island, Nebraska
  - Investigational Site Number 840015, Omaha, Nebraska
  - Investigational Site Number 840021, Omaha, Nebraska
  - Investigational Site Number 840001, Omaha, Nebraska
  - Investigational Site Number 840221, Las Vegas, Nevada
  - Investigational Site Number 840062, Nashua, New Hampshire
  - Investigational Site Number 840077, Bridgewater, New Jersey
  - Investigational Site Number 840173, Bridgewater, New Jersey
  - Investigational Site Number 840127, Flemington, New Jersey
  - Investigational Site Number 840359, Hackensack, New Jersey
  - Investigational Site Number 840348, Moorestown, New Jersey
  - Investigational Site Number 840128, New Brunswick, New Jersey
  - Investigational Site Number 840167, Pomona, New Jersey
  - Investigational Site Number 840067, Ridgewood, New Jersey
  - Investigational Site Number 840250, Somerset, New Jersey
  - Investigational Site Number 840277, Voorhees Township, New Jersey
  - Investigational Site Number 840083, Westwood, New Jersey
  - Investigational Site Number 840322, Buffalo, New York
  - Investigational Site Number 840248, New York, New York
  - Investigational Site Number 840371, New York, New York
  - Investigational Site Number 840333, Newburgh, New York
  - Investigational Site Number 840017, Poughkeepsie, New York
  - Investigational Site Number 840222, The Bronx, New York
  - Investigational Site Number 840166, Valhalla, New York
  - Investigational Site Number 840354, Williamsville, New York
  - Investigational Site Number 840070, Elizabeth City, North Carolina
  - Investigational Site Number 840303, Greenville, North Carolina
  - Investigational Site Number 840182, Greenville, North Carolina
  - Investigational Site Number 840243, Raleigh, North Carolina
  - Investigational Site Number 840342, Raleigh, North Carolina
  - Investigational Site Number 840293, Rocky Mount, North Carolina
  - Investigational Site Number 840088, Statesville, North Carolina
  - Investigational Site Number 840052, Wilmington, North Carolina
  - Investigational Site Number 840214, Fargo, North Dakota
  - Investigational Site Number 840306, Glasston, North Dakota
  - Investigational Site Number 840095, Minot, North Dakota
  - Investigational Site Number 840257, Mountain Lakes, North Dakota
  - Investigational Site Number 840364, Akron, Ohio
  - Investigational Site Number 840131, Cincinnati, Ohio
  - Investigational Site Number 840045, Columbus, Ohio
  - Investigational Site Number 840265, Columbus, Ohio
  - Investigational Site Number 840113, Lorain, Ohio
  - Investigational Site Number 840115, Lorain, Ohio
  - Investigational Site Number 840309, Maumee, Ohio
  - Investigational Site Number 840297, Springfield, Ohio
  - Investigational Site Number 840172, Toledo, Ohio
  - Investigational Site Number 840263, Youngstown, Ohio
  - Investigational Site Number 840334, Oklahoma City, Oklahoma
  - Investigational Site Number 840337, Oklahoma City, Oklahoma
  - Investigational Site Number 840018, Tulsa, Oklahoma
  - Investigational Site Number 840184, Portland, Oregon
  - Investigational Site Number 840133, Allentown, Pennsylvania
  - Investigational Site Number 840104, Beaver, Pennsylvania
  - Investigational Site Number 840170, Camp Hill, Pennsylvania
  - Investigational Site Number 840020, Doylestown, Pennsylvania
  - Investigational Site Number 840016, Erie, Pennsylvania
  - Investigational Site Number 840329, Goodyear, Pennsylvania
  - Investigational Site Number 840126, Knoxville, Pennsylvania
  - Investigational Site Number 840249, Lancaster, Pennsylvania
  - Investigational Site Number 840150, Lancaster, Pennsylvania
  - Investigational Site Number 840231, Philadelphia, Pennsylvania
  - Investigational Site Number 840339, Philadelphia, Pennsylvania
  - Investigational Site Number 840230, Pittsburgh, Pennsylvania
  - Investigational Site Number 840028, Sayre, Pennsylvania
  - Investigational Site Number 840069, Scranton, Pennsylvania
  - Investigational Site Number 840316, Scranton, Pennsylvania
  - Investigational Site Number 840273, Seven Fields, Pennsylvania
  - Investigational Site Number 840227, Washington, Pennsylvania
  - Investigational Site Number 840129, Pawtucket, Rhode Island
  - Investigational Site Number 840118, Anderson, South Carolina
  - Investigational Site Number 840190, Greenwood, South Carolina
  - Investigational Site Number 840360, Lancaster, South Carolina
  - Investigational Site Number 840314, Myrtle Beach, South Carolina
  - Investigational Site Number 840008, Rapid City, South Dakota
  - Investigational Site Number 840285, Chattanooga, Tennessee
  - Investigational Site Number 840287, Jackson, Tennessee
  - Investigational Site Number 840040, Johnson City, Tennessee
  - Investigational Site Number 840238, Knoxville, Tennessee
  - Investigational Site Number 840195, Oak Ridge, Tennessee
  - Investigational Site Number 840205, Amarillo, Texas
  - Investigational Site Number 840352, Amarillo, Texas
  - Investigational Site Number 840135, Austin, Texas
  - Investigational Site Number 840301, Dallas, Texas
  - Investigational Site Number 840152, Dallas, Texas
  - Investigational Site Number 840157, Dallas, Texas
  - Investigational Site Number 840229, Fort Worth, Texas
  - Investigational Site Number 840120, Fort Worth, Texas
  - Investigational Site Number 840258, Fort Worth, Texas
  - Investigational Site Number 840136, Kingwood, Texas
  - Investigational Site Number 840027, Lubbock, Texas
  - Investigational Site Number 840202, Lufkin, Texas
  - Investigational Site Number 840270, Odessa, Texas
  - Investigational Site Number 840162, San Antonio, Texas
  - Investigational Site Number 840232, San Antonio, Texas
  - Investigational Site Number 840328, Schertz, Texas
  - Investigational Site Number 840158, Tyler, Texas
  - Investigational Site Number 840318, Victoria, Texas
  - Investigational Site Number 840245, Wichita Falls, Texas
  - Investigational Site Number 840256, Orem, Utah
  - Investigational Site Number 840296, Salt Lake City, Utah
  - Investigational Site Number 840053, Burlington, Vermont
  - Investigational Site Number 840049, Charlottesville, Virginia
  - Investigational Site Number 840260, Charlottesville, Virginia
  - Investigational Site Number 840350, Harrisonburg, Virginia
  - Investigational Site Number 840215, Leesburg, Virginia
  - Investigational Site Number 840010, Lynchburg, Virginia
  - Investigational Site Number 840225, Manassas, Virginia
  - Investigational Site Number 840022, Richmond, Virginia
  - Investigational Site Number 840078, Richmond, Virginia
  - Investigational Site Number 840110, Richmond, Virginia
  - Investigational Site Number 840149, Roanoke, Virginia
  - Investigational Site Number 840223, Winchester, Virginia
  - Investigational Site Number 840025, Bellevue, Washington
  - Investigational Site Number 840321, Everett, Washington
  - Investigational Site Number 840326, Spokane, Washington
  - Investigational Site Number 840086, Tacoma, Washington
  - Investigational Site Number 840295, Walla Walla, Washington
  - Investigational Site Number 840262, Burlington, Wisconsin
  - Investigational Site Number 840298, Green Bay, Wisconsin
  - Investigational Site Number 840059, Green Bay, Wisconsin
  - Investigational Site Number 840177, La Crosse, Wisconsin
  - Investigational Site Number 840300, Manitowoc, Wisconsin
- Argentina (52):
  - Investigational Site Number 032012, Adrogué
  - Investigational Site Number 032018, Bahía Blanca
  - Investigational Site Number 032050, Caba
  - Investigational Site Number 032048, Caba
  - Investigational Site Number 032023, Caba
  - Investigational Site Number 032020, Caba
  - Investigational Site Number 032041, Caba
  - Investigational Site Number 032011, Caba
  - Investigational Site Number 032045, Caba
  - Investigational Site Number 032010, Ciudad de Buenos Aires
  - Investigational Site Number 032046, Ciudadela
  - Investigational Site Number 032017, Coronel Suárez
  - Investigational Site Number 032009, Corrientes
  - Investigational Site Number 032032, Córdoba
  - Investigational Site Number 032019, Córdoba
  - Investigational Site Number 032021, Córdoba
  - Investigational Site Number 032026, Córdoba
  - Investigational Site Number 032008, Córdoba
  - Investigational Site Number 032049, Córdoba
  - Investigational Site Number 032042, Córdoba
  - Investigational Site Number 032038, Córdoba
  - Investigational Site Number 032031, Córdoba
  - Investigational Site Number 032005, Junín
  - Investigational Site Number 032001, La Plata
  - Investigational Site Number 032040, La Plata
  - Investigational Site Number 032033, Mar del Plata
  - Investigational Site Number 032014, Mar del Plata
  - Investigational Site Number 032016, Mendoza
  - Investigational Site Number 032030, Merlo
  - Investigational Site Number 032036, Morón
  - Investigational Site Number 032007, Olivos
  - Investigational Site Number 032044, Olivos
  - Investigational Site Number 032004, Quilmes
  - Investigational Site Number 032025, Rafaela
  - Investigational Site Number 032035, Ramos Mejía
  - Investigational Site Number 032039, Resistencia
  - Investigational Site Number 032028, Rosario
  - Investigational Site Number 032024, Rosario
  - Investigational Site Number 032053, Salta
  - Investigational Site Number 032037, San Isidro
  - Investigational Site Number 032052, San Martín
  - Investigational Site Number 032013, San Martín
  - Investigational Site Number 032002, San Miguel de Tucumán
  - Investigational Site Number 032034, San Miguel de Tucumán
  - Investigational Site Number 032006, San Nicolás
  - Investigational Site Number 032043, Santa Fe
  - Investigational Site Number 032003, Santa Fe
  - Investigational Site Number 032051, Santa Rosa
  - Investigational Site Number 032047, Santiago del Estero
  - Investigational Site Number 032029, Venado Tuerto
  - Investigational Site Number 032022, Villa María
  - Investigational Site Number 032015, Zárate
- Australia (25):
  - Investigational Site Number 036002, Ashford
  - Investigational Site Number 036023, Auchenflower
  - Investigational Site Number 036024, Ballarat
  - Investigational Site Number 036020, Bedford Park
  - Investigational Site Number 036015, Bruce
  - Investigational Site Number 036026, Cairns
  - Investigational Site Number 036005, Chermside
  - Investigational Site Number 036008, Chermside
  - Investigational Site Number 036011, Coffs Harbour
  - Investigational Site Number 036003, Concord
  - Investigational Site Number 036017, Elizabeth Vale
  - Investigational Site Number 036006, Fullarton
  - Investigational Site Number 036004, Gosford
  - Investigational Site Number 036019, Heidelberg West
  - Investigational Site Number 036027, Hobart
  - Investigational Site Number 036009, Kogarah
  - Investigational Site Number 036012, Mildura
  - Investigational Site Number 036028, Nambour
  - Investigational Site Number 036013, New Lambton
  - Investigational Site Number 036010, Perth
  - Investigational Site Number 036014, Prahran
  - Investigational Site Number 036018, Redcliffe
  - Investigational Site Number 036022, Richmond
  - Investigational Site Number 036025, Woodville South
  - Investigational Site Number 036021, Woolloongabba
- Austria (6):
  - Investigational Site Number 040004, Feldkirch
  - Investigational Site Number 040007, Graz
  - Investigational Site Number 040001, Salzburg
  - Investigational Site Number 040006, Vienna
  - Investigational Site Number 040003, Vienna
  - Investigational Site Number 040002, Vienna
- Belgium (21):
  - Investigational Site Number 056016, Aalst
  - Investigational Site Number 056003, Antwerp
  - Investigational Site Number 056002, Antwerp
  - Investigational Site Number 056008, Bonheiden
  - Investigational Site Number 056014, Brasschaat
  - Investigational Site Number 056005, Brussels
  - Investigational Site Number 056021, Brussels
  - Investigational Site Number 056004, Brussels
  - Investigational Site Number 056017, Edegem
  - Investigational Site Number 056024, Genk
  - Investigational Site Number 056007, Ghent
  - Investigational Site Number 056018, Ghent
  - Investigational Site Number 056020, La Louvière
  - Investigational Site Number 056009, Leuven
  - Investigational Site Number 056015, Liège
  - Investigational Site Number 056010, Mechelen
  - Investigational Site Number 056013, Mol
  - Investigational Site Number 056001, Ottignies
  - Investigational Site Number 056012, Overpelt
  - Investigational Site Number 056006, Roeselare
  - Investigational Site Number 056019, Tienen
- Bosnia and Herzegovina (11):
  - Investigational Site Number 070001, Banja Luka
  - Investigational Site Number 070002, Banja Luka
  - Investigational Site Number 070011, Bihać
  - Investigational Site Number 070003, Mostar
  - Investigational Site Number 070004, Mostar
  - Investigational Site Number 070005, Sarajevo
  - Investigational Site Number 070007, Sarajevo
  - Investigational Site Number 070010, Sarajevo
  - Investigational Site Number 070008, Tuzla
  - Investigational Site Number 070009, Tuzla
  - Investigational Site Number 070006, Zenica
- Brazil (41):
  - Investigational Site Number 076029, Aparecida de Goiânia
  - Investigational Site Number 076032, Belém
  - Investigational Site Number 076017, Belo Horizonte
  - Investigational Site Number 076004, Belo Horizonte
  - Investigational Site Number 076022, Belo Horizonte
  - Investigational Site Number 076038, Belo Horizonte
  - Investigational Site Number 076002, Blumenau
  - Investigational Site Number 076011, Brasília
  - Investigational Site Number 076007, Brasília
  - Investigational Site Number 076003, Campina Grande do Sul
  - Investigational Site Number 076006, Campinas
  - Investigational Site Number 076040, Canoas
  - Investigational Site Number 076033, Curitiba
  - Investigational Site Number 076005, Curitiba
  - Investigational Site Number 076009, Fortaleza
  - Investigational Site Number 076008, Fortaleza
  - Investigational Site Number 076012, Goiânia
  - Investigational Site Number 076021, Goiânia
  - Investigational Site Number 076019, Passo Fundo
  - Investigational Site Number 076018, Pelotas
  - Investigational Site Number 076024, Porto Alegre
  - Investigational Site Number 076026, Porto Alegre
  - Investigational Site Number 076014, Porto Alegre
  - Investigational Site Number 076001, Porto Alegre
  - Investigational Site Number 076027, Porto Alegre
  - Investigational Site Number 076035, Riberao Preto
  - Investigational Site Number 076010, Rio de Janeiro
  - Investigational Site Number 076015, Salvador
  - Investigational Site Number 076041, Salvador
  - Investigational Site Number 076036, Santo André
  - Investigational Site Number 076031, São Bernardo do Campo
  - Investigational Site Number 076030, São José do Rio Preto
  - Investigational Site Number 076020, São José do Rio Preto
  - Investigational Site Number 076025, São Paulo
  - Investigational Site Number 076042, São Paulo
  - Investigational Site Number 076039, São Paulo
  - Investigational Site Number 076013, São Paulo
  - Investigational Site Number 076023, São Paulo
  - Investigational Site Number 076028, São Paulo
  - Investigational Site Number 076016, Tatuí
  - Investigational Site Number 076034, Uberlândia
- Bulgaria (18):
  - Investigational Site Number 100020, Blagoevgrad
  - Investigational Site Number 100012, Burgas
  - Investigational Site Number 100011, Pazardzhik
  - Investigational Site Number 100013, Pleven
  - Investigational Site Number 100018, Pleven
  - Investigational Site Number 100005, Plovdiv
  - Investigational Site Number 100015, Sandanski
  - Investigational Site Number 100023, Smolyan
  - Investigational Site Number 100017, Sofia
  - Investigational Site Number 100007, Sofia
  - Investigational Site Number 100001, Sofia
  - Investigational Site Number 100004, Sofia
  - Investigational Site Number 100010, Sofia
  - Investigational Site Number 100019, Sofia
  - Investigational Site Number 100016, Sofia
  - Investigational Site Number 100003, Sofia
  - Investigational Site Number 100022, Varna
  - Investigational Site Number 100014, Veliko Tarnovo
- Canada (42):
  - Investigational Site Number 124033, Calgary
  - Investigational Site Number 124017, Cambridge
  - Investigational Site Number 124013, Cambridge
  - Investigational Site Number 124026, Edmonton
  - Investigational Site Number 124019, Edmonton
  - Investigational Site Number 124016, Edmonton
  - Investigational Site Number 124027, Granby
  - Investigational Site Number 124002, Halifax
  - Investigational Site Number 124051, Hamilton
  - Investigational Site Number 124043, Joliette
  - Investigational Site Number 124045, Kitchener
  - Investigational Site Number 124053, Lévis
  - Investigational Site Number 124015, Longueuil
  - Investigational Site Number 124004, Moncton
  - Investigational Site Number 124040, Montreal
  - Investigational Site Number 124032, Montreal
  - Investigational Site Number 124036, Montreal
  - Investigational Site Number 124042, Montreal
  - Investigational Site Number 124028, New Westminster
  - Investigational Site Number 124008, Newmarket
  - Investigational Site Number 124005, Oshawa
  - Investigational Site Number 124007, Ottawa
  - Investigational Site Number 124006, Penticton
  - Investigational Site Number 124012, Red Deer
  - Investigational Site Number 124054, Saint-Jérôme
  - Investigational Site Number 124024, Sainte-Foy
  - Investigational Site Number 124035, Scarborough
  - Investigational Site Number 124047, Sherbrooke
  - Investigational Site Number 124044, St. Catherines
  - Investigational Site Number 124025, St. Georges
  - Investigational Site Number 124034, St. John's
  - Investigational Site Number 124021, St. John's
  - Investigational Site Number 124009, Surrey
  - Investigational Site Number 124022, Sydney
  - Investigational Site Number 124048, Thetford-Mines
  - Investigational Site Number 124037, Thunder Bay
  - Investigational Site Number 124001, Toronto
  - Investigational Site Number 124049, Trois-Rivières
  - Investigational Site Number 124039, Vancouver
  - Investigational Site Number 124023, Victoria
  - Investigational Site Number 124041, Victoria
  - Investigational Site Number 124038, Winnipeg
- Chile (18):
  - Investigational Site Number 152013, Concepción
  - Investigational Site Number 152003, Osorno
  - Investigational Site Number 152017, Punta Arenas
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152014, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152019, Santiago
  - Investigational Site Number 152007, Santiago
  - Investigational Site Number 152012, Santiago
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152006, Santiago
  - Investigational Site Number 152016, Santiago
  - Investigational Site Number 152015, Santiago
  - Investigational Site Number 152009, Talca
  - Investigational Site Number 152002, Temuco
  - Investigational Site Number 152008, Valdivia
  - Investigational Site Number 152010, Viña del Mar
  - Investigational Site Number 152018, Viña del Mar
- China (63):
  - Investigational Site Number 156022, Baotou
  - Investigational Site Number 156004, Beijing
  - Investigational Site Number 156005, Beijing
  - Investigational Site Number 156006, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156082, Beijing
  - Investigational Site Number 156009, Beijing
  - Investigational Site Number 156003, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156013, Changchun
  - Investigational Site Number 156064, Changchun
  - Investigational Site Number 156052, Changsha
  - Investigational Site Number 156053, Changsha
  - Investigational Site Number 156088, Changsha
  - Investigational Site Number 156057, Chongqing
  - Investigational Site Number 156070, Fuzhou
  - Investigational Site Number 156079, Fuzhou
  - Investigational Site Number 156059, Guangzhou
  - Investigational Site Number 156060, Guangzhou
  - Investigational Site Number 156071, Guangzhou
  - Investigational Site Number 156061, Guangzhou
  - Investigational Site Number 156072, Guiyang
  - Investigational Site Number 156047, Hangzhou
  - Investigational Site Number 156077, Hangzhou
  - Investigational Site Number 156048, Hangzhou
  - Investigational Site Number 156068, Hangzhou
  - Investigational Site Number 156078, Hangzhou
  - Investigational Site Number 156046, Hangzhou
  - Investigational Site Number 156020, Hohhot
  - Investigational Site Number 156032, Jinan
  - Investigational Site Number 156031, Jinan
  - Investigational Site Number 156027, Lanzhou
  - Investigational Site Number 156074, Lanzhou
  - Investigational Site Number 156081, Luzhou
  - Investigational Site Number 156054, Nanchang
  - Investigational Site Number 156055, Nanchang
  - Investigational Site Number 156034, Nanjing
  - Investigational Site Number 156035, Nanjing
  - Investigational Site Number 156039, Shanghai
  - Investigational Site Number 156076, Shanghai
  - Investigational Site Number 156044, Shanghai
  - Investigational Site Number 156043, Shanghai
  - Investigational Site Number 156038, Shanghai
  - Investigational Site Number 156040, Shanghai
  - Investigational Site Number 156016, Shenyang
  - Investigational Site Number 156017, Shenyang
  - Investigational Site Number 156073, Shenzhen
  - Investigational Site Number 156084, Shenzhen
  - Investigational Site Number 156063, Siping
  - Investigational Site Number 156037, Suzhou
  - Investigational Site Number 156066, Tianjin
  - Investigational Site Number 156067, Tianjin
  - Investigational Site Number 156083, Tianjin
  - Investigational Site Number 156025, Tianjin
  - Investigational Site Number 156065, Wenzhou
  - Investigational Site Number 156051, Wuhan
  - Investigational Site Number 156087, Wuhan
  - Investigational Site Number 156029, Xi'an
  - Investigational Site Number 156086, Xi'an
  - Investigational Site Number 156062, Xuzhou
  - Investigational Site Number 156014, Yanji
  - Investigational Site Number 156075, Yueyang
  - Investigational Site Number 156080, Zhanjiang
- Colombia (17):
  - Investigational Site Number 170006, Armenia
  - Investigational Site Number 170003, Barranquilla
  - Investigational Site Number 170011, Barranquilla
  - Investigational Site Number 170013, Barranquilla
  - Investigational Site Number 170022, Bogota D.C.
  - Investigational Site Number 170018, Bogotá
  - Investigational Site Number 170016, Bogotá
  - Investigational Site Number 170010, Cali
  - Investigational Site Number 170001, Cali
  - Investigational Site Number 170017, Cartagena
  - Investigational Site Number 170004, Cartagena
  - Investigational Site Number 170008, Espinal - Tolima
  - Investigational Site Number 170005, Floridablanca
  - Investigational Site Number 170002, Manizales
  - Investigational Site Number 170007, Medellín
  - Investigational Site Number 170009, Medellín
  - Investigational Site Number 170021, Medellín
- Croatia (16):
  - Investigational Site Number 191013, Dubrovnik
  - Investigational Site Number 191017, Krapinske Toplice
  - Investigational Site Number 191009, Opatija
  - Investigational Site Number 191006, Rijeka
  - Investigational Site Number 191012, Slavonski Brod
  - Investigational Site Number 191003, Varaždin
  - Investigational Site Number 191001, Zagreb
  - Investigational Site Number 191002, Zagreb
  - Investigational Site Number 191005, Zagreb
  - Investigational Site Number 191007, Zagreb
  - Investigational Site Number 191008, Zagreb
  - Investigational Site Number 191010, Zagreb
  - Investigational Site Number 191011, Zagreb
  - Investigational Site Number 191015, Zagreb
  - Investigational Site Number 191016, Zagreb
  - Investigational Site Number 191018, Zagreb
- Czechia (22):
  - Investigational Site Number 203003, Brno
  - Investigational Site Number 203020, Česká Lípa
  - Investigational Site Number 203025, Český Krumlov
  - Investigational Site Number 203023, Hodonín
  - Investigational Site Number 203006, Hradec Králové
  - Investigational Site Number 203019, Kladno
  - Investigational Site Number 203005, Kladno
  - Investigational Site Number 203008, Kroměříž
  - Investigational Site Number 203015, Liberec
  - Investigational Site Number 203024, Mariánské Lázně
  - Investigational Site Number 203013, Olomouc
  - Investigational Site Number 203016, Ostrava
  - Investigational Site Number 203014, Pardubice
  - Investigational Site Number 203018, Pilsen
  - Investigational Site Number 203011, Prague
  - Investigational Site Number 203017, Prague
  - Investigational Site Number 203004, Prague
  - Investigational Site Number 203021, Prague
  - Investigational Site Number 203012, Prague
  - Investigational Site Number 203007, Praha 5 - Motol
  - Investigational Site Number 203009, Rakovník
  - Investigational Site Number 203010, Zlín
- Denmark (17):
  - Investigational Site Number 208016, Aabenraa
  - Investigational Site Number 208012, Aalborg
  - Investigational Site Number 208011, Aarhus N
  - Investigational Site Number 208002, Copenhagen
  - Investigational Site Number 208003, Glostrup Municipality
  - Investigational Site Number 208007, Hellerup
  - Investigational Site Number 208006, Herning
  - Investigational Site Number 208018, Hillerød
  - Investigational Site Number 208014, Holbæk
  - Investigational Site Number 208013, Hvidovre
  - Investigational Site Number 208004, Køge
  - Investigational Site Number 208017, Næstved
  - Investigational Site Number 208009, Odense C
  - Investigational Site Number 208015, Silkeborg
  - Investigational Site Number 208008, Slagelse
  - Investigational Site Number 208001, Vejle
  - Investigational Site Number 208010, Viborg
- Estonia (7):
  - Investigational Site Number 233007, Pärnu
  - Investigational Site Number 233004, Tallinn
  - Investigational Site Number 233002, Tallinn
  - Investigational Site Number 233001, Tallinn
  - Investigational Site Number 233005, Tallinn
  - Investigational Site Number 233003, Tartu
  - Investigational Site Number 233006, Viljandimaa
- Finland (4):
  - Investigational Site Number 246004, Helsinki
  - Investigational Site Number 246001, Oulu
  - Investigational Site Number 246003, Tampere
  - Investigational Site Number 246002, Turku
- France (22):
  - Investigational Site Number 250003, Besançon
  - Investigational Site Number 250007, Brest
  - Investigational Site Number 250010, Cambrai
  - Investigational Site Number 250018, Clermont-Ferrand
  - Investigational Site Number 250021, Compiègne
  - Investigational Site Number 250002, Dijon
  - Investigational Site Number 250001, Grenoble
  - Investigational Site Number 250009, Limoges
  - Investigational Site Number 250019, Marseille
  - Investigational Site Number 250008, Massy
  - Investigational Site Number 250005, Montfermeil
  - Investigational Site Number 250023, Montpellier
  - Investigational Site Number 250025, Nantes
  - Investigational Site Number 250017, Nice
  - Investigational Site Number 250020, Paris
  - Investigational Site Number 250012, Paris
  - Investigational Site Number 250004, Paris
  - Investigational Site Number 250015, Paris
  - Investigational Site Number 250011, Pau
  - Investigational Site Number 250016, Pessac
  - Investigational Site Number 250026, Rouen
  - Investigational Site Number 250022, Strasbourg
- Georgia (7):
  - Investigational Site Number 268004, Batumi
  - Investigational Site Number 268001, Kutaisi
  - Investigational Site Number 268005, Tbilisi
  - Investigational Site Number 268002, Tbilisi
  - Investigational Site Number 268003, Tbilisi
  - Investigational Site Number 268008, Tbilisi
  - Investigational Site Number 268009, Tbilisi
- Germany (42):
  - Investigational Site Number 276013, Aachen
  - Investigational Site Number 276019, Bad Krozingen
  - Investigational Site Number 276008, Berlin
  - Investigational Site Number 276040, Berlin
  - Investigational Site Number 276051, Berlin
  - Investigational Site Number 276039, Berlin
  - Investigational Site Number 276025, Berlin
  - Investigational Site Number 276054, Bernau
  - Investigational Site Number 276037, Bielefeld
  - Investigational Site Number 276016, Bonn
  - Investigational Site Number 276009, Bonn
  - Investigational Site Number 276001, Dortmund
  - Investigational Site Number 276006, Dortmund
  - Investigational Site Number 276031, Dortmund
  - Investigational Site Number 276050, Dresden
  - Investigational Site Number 276024, Eschweiler
  - Investigational Site Number 276028, Essen
  - Investigational Site Number 276036, Frankfurt am Main
  - Investigational Site Number 276012, Freiburg im Breisgau
  - Investigational Site Number 276030, Halle
  - Investigational Site Number 276032, Hamburg
  - Investigational Site Number 276017, Hamburg
  - Investigational Site Number 276027, Hamburg
  - Investigational Site Number 276029, Hamm
  - Investigational Site Number 276052, Haßloch
  - Investigational Site Number 276014, Heidelberg
  - Investigational Site Number 276023, Homburg/Saar
  - Investigational Site Number 276035, Kassel
  - Investigational Site Number 276046, Leipzig
  - Investigational Site Number 276020, Limburg
  - Investigational Site Number 276026, Lippstadt
  - Investigational Site Number 276044, Lübeck
  - Investigational Site Number 276021, Magdeburg
  - Investigational Site Number 276015, Mainz
  - Investigational Site Number 276010, Marburg
  - Investigational Site Number 276018, Münster
  - Investigational Site Number 276042, Nuremberg
  - Investigational Site Number 276048, Peine
  - Investigational Site Number 276053, Rotenburg an der Fulda
  - Investigational Site Number 276045, Rüdersdorf Bei Berlin
  - Investigational Site Number 276002, Stuttgart
  - Investigational Site Number 276033, Warendorf
- Greece (12):
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300002, Athens
  - Investigational Site Number 300007, Athens
  - Investigational Site Number 300008, Chios
  - Investigational Site Number 300013, Haidari
  - Investigational Site Number 300010, Heraklion
  - Investigational Site Number 300005, Ioannina
  - Investigational Site Number 300003, Marousi
  - Investigational Site Number 300006, N. Ionia
  - Investigational Site Number 300004, Pátrai
  - Investigational Site Number 300011, Thessaloniki
  - Investigational Site Number 300009, Thessaloniki
- Guatemala (4):
  - Investigational Site Number 320003, Guatemala City
  - Investigational Site Number 320001, Guatemala City
  - Investigational Site Number 320002, Guatemala City
  - Investigational Site Number 320004, Guatemala City
- Hong Kong (2):
  - Investigational Site Number 344003, Hong Kong
  - Investigational Site Number 344001, Shatin, Nt
- Hungary (13):
  - Investigational Site Number 348013, Balatonfüred
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348012, Budapest
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348008, Debrecen
  - Investigational Site Number 348004, Eger
  - Investigational Site Number 348003, Gyula
  - Investigational Site Number 348010, Pécs
  - Investigational Site Number 348009, Szeged
  - Investigational Site Number 348007, Székesfehérvár
  - Investigational Site Number 348011, Szombathely
  - Investigational Site Number 348001, Zalaegerszeg
- India (56):
  - Investigational Site Number 356060, Ahmedabad
  - Investigational Site Number 356056, Aurangabad
  - Investigational Site Number 356025, Bangalore
  - Investigational Site Number 356028, Bangalore
  - Investigational Site Number 356083, Bangalore
  - Investigational Site Number 356018, Bangalore
  - Investigational Site Number 356026, Bangalore
  - Investigational Site Number 356084, Bangalore
  - Investigational Site Number 356103, Belagavi
  - Investigational Site Number 356019, Bikaner
  - Investigational Site Number 356013, Chennai
  - Investigational Site Number 356012, Chennai
  - Investigational Site Number 356081, Chennai
  - Investigational Site Number 356093, Delhi
  - Investigational Site Number 356038, Delhi
  - Investigational Site Number 356101, Gūrgaon
  - Investigational Site Number 356100, Gūrgaon
  - Investigational Site Number 356035, Hyderabad
  - Investigational Site Number 356082, Hyderabad
  - Investigational Site Number 356015, Jaipur
  - Investigational Site Number 356053, Karad
  - Investigational Site Number 356102, Karamsad
  - Investigational Site Number 356022, Kochi
  - Investigational Site Number 356106, Kolhāpur
  - Investigational Site Number 356067, Kolkata
  - Investigational Site Number 356079, Kolkata
  - Investigational Site Number 356069, Kolkata
  - Investigational Site Number 356089, Ludhiana
  - Investigational Site Number 356095, Mangalore
  - Investigational Site Number 356071, Mumbai
  - Investigational Site Number 356057, Mumbai
  - Investigational Site Number 356007, Mysore
  - Investigational Site Number 356087, Nagpur
  - Investigational Site Number 356098, Nagpur
  - Investigational Site Number 356097, Nagpur
  - Investigational Site Number 356096, Nashik
  - Investigational Site Number 356055, New Delhi
  - Investigational Site Number 356031, New Delhi
  - Investigational Site Number 356041, Panjim
  - Investigational Site Number 356077, Pune
  - Investigational Site Number 356099, Pune
  - Investigational Site Number 356048, Pune
  - Investigational Site Number 356049, Pune
  - Investigational Site Number 356050, Pune
  - Investigational Site Number 356045, Pune
  - Investigational Site Number 356046, Pune
  - Investigational Site Number 356094, Pune
  - Investigational Site Number 356009, Secunderabad
  - Investigational Site Number 356032, Secunderabad
  - Investigational Site Number 356042, Secunderabad, Hyderabad
  - Investigational Site Number 356091, Surat
  - Investigational Site Number 356002, Vijayawada
  - Investigational Site Number 356105, Vijaywada
  - Investigational Site Number 356033, Visakhapatnam
  - Investigational Site Number 356039, Vishkhapattanam
  - Investigational Site Number 356104, Wardha
- Israel (27):
  - Investigational Site Number 376006, Afula
  - Investigational Site Number 376024, Afula
  - Investigational Site Number 376009, Ashkelon
  - Investigational Site Number 376012, Beersheba
  - Investigational Site Number 376011, Haifa
  - Investigational Site Number 376017, Haifa
  - Investigational Site Number 376025, Haifa
  - Investigational Site Number 376018, Haifa
  - Investigational Site Number 376007, Holon
  - Investigational Site Number 376021, Holon
  - Investigational Site Number 376016, Jerusalem
  - Investigational Site Number 376005, Jerusalem
  - Investigational Site Number 376027, Jerusalem
  - Investigational Site Number 376002, Kfar Saba
  - Investigational Site Number 376013, Kfar Saba
  - Investigational Site Number 376004, Nahariya
  - Investigational Site Number 376015, Nazareth
  - Investigational Site Number 376001, Petah Tikva
  - Investigational Site Number 376019, Petah Tikva
  - Investigational Site Number 376020, Rehovot
  - Investigational Site Number 376003, Safed
  - Investigational Site Number 376008, Safed
  - Investigational Site Number 376010, Tel Aviv
  - Investigational Site Number 376014, Tel Aviv
  - Investigational Site Number 376022, Tel Litwinsky
  - Investigational Site Number 376023, Tiberias
  - Investigational Site Number 376026, Tzrifin
- Italy (24):
  - Investigational Site Number 380019, Augusta
  - Investigational Site Number 380017, Bergamo
  - Investigational Site Number 380026, Brescia
  - Investigational Site Number 380008, Brescia
  - Investigational Site Number 380012, Ferrara
  - Investigational Site Number 380027, Forlì
  - Investigational Site Number 380015, Livorno
  - Investigational Site Number 380033, Massa
  - Investigational Site Number 380030, Milan
  - Investigational Site Number 380005, Milan
  - Investigational Site Number 380003, Milan
  - Investigational Site Number 380025, Monza
  - Investigational Site Number 380001, Napoli
  - Investigational Site Number 380002, Napoli
  - Investigational Site Number 380021, Novara
  - Investigational Site Number 380009, Osio Sotto
  - Investigational Site Number 380007, Palermo
  - Investigational Site Number 380013, Perugia
  - Investigational Site Number 380031, Rho
  - Investigational Site Number 380014, Rimini
  - Investigational Site Number 380024, Roma
  - Investigational Site Number 380028, Seriate
  - Investigational Site Number 380032, Treviso
  - Investigational Site Number 380020, Vittorio Veneto
- Japan (39):
  - Investigational Site Number 392013, Amagasaki-Shi
  - Investigational Site Number 392041, Amagasaki-Shi
  - Investigational Site Number 392029, Fukuoka
  - Investigational Site Number 392019, Hachioji-Shi
  - Investigational Site Number 392026, Higashihiroshima-Shi
  - Investigational Site Number 392024, Higashiibaraki-Gun
  - Investigational Site Number 392003, Hiroshima
  - Investigational Site Number 392002, Itabashi-Ku
  - Investigational Site Number 392014, Itabashi-Ku
  - Investigational Site Number 392033, Izumisano
  - Investigational Site Number 392020, Kanazawa
  - Investigational Site Number 392015, Kitakyushu-Shi
  - Investigational Site Number 392017, Kobe
  - Investigational Site Number 392028, Kobe
  - Investigational Site Number 392037, Kobe
  - Investigational Site Number 392025, Koga-Shi
  - Investigational Site Number 392010, Komatsu-Shi
  - Investigational Site Number 392035, Komatsushima-Shi
  - Investigational Site Number 392023, Kumamoto
  - Investigational Site Number 392031, Kumamoto
  - Investigational Site Number 392039, Kure-Shi
  - Investigational Site Number 392012, Kurume-Shi
  - Investigational Site Number 392032, Kusatsu-Shi
  - Investigational Site Number 392001, Kyoto
  - Investigational Site Number 392027, Minatoku
  - Investigational Site Number 392016, Morioka
  - Investigational Site Number 392005, Nagoya
  - Investigational Site Number 392022, Nerima-Ku
  - Investigational Site Number 392009, Osaka
  - Investigational Site Number 392011, Osaka
  - Investigational Site Number 392040, Osaka
  - Investigational Site Number 392004, Sagamihara-Shi
  - Investigational Site Number 392036, Sapporo
  - Investigational Site Number 392034, Shinagawa-Ku
  - Investigational Site Number 392018, Suita-Shi
  - Investigational Site Number 392030, Tokushima
  - Investigational Site Number 392008, Urasoe-Shi
  - Investigational Site Number 392006, Yokohama
  - Investigational Site Number 392021, Yokohama
- Latvia (6):
  - Investigational Site Number 428004, Daugavpils
  - Investigational Site Number 428002, Liepāja
  - Investigational Site Number 428006, Riga
  - Investigational Site Number 428001, Riga
  - Investigational Site Number 428005, Riga
  - Investigational Site Number 428003, Ventspils
- Lithuania (9):
  - Investigational Site Number 440004, Kaunas
  - Investigational Site Number 440005, Kaunas
  - Investigational Site Number 440009, Kaunas
  - Investigational Site Number 440008, Kaunas
  - Investigational Site Number 440001, Klaipėda
  - Investigational Site Number 440006, Klaipėda
  - Investigational Site Number 440002, Vilnius
  - Investigational Site Number 440007, Vilnius
  - Investigational Site Number 440003, Vilnius
- Malaysia (7):
  - Investigational Site Number 458004, Batu Caves
  - Investigational Site Number 458007, Kota Bharu
  - Investigational Site Number 458006, Kota Kinabalu
  - Investigational Site Number 458002, Kuala Lumpur
  - Investigational Site Number 458005, Kuala Lumpur
  - Investigational Site Number 458003, Kuching
  - Investigational Site Number 458001, Sungai Buloh
- Mexico (20):
  - Investigational Site Number 484005, Aguascalientes
  - Investigational Site Number 484015, Aguascalientes
  - Investigational Site Number 484004, Culiacán
  - Investigational Site Number 484003, Durango
  - Investigational Site Number 484010, Guadalajara
  - Investigational Site Number 484006, Guadalajara
  - Investigational Site Number 484008, Jalapa
  - Investigational Site Number 484023, Mexico City
  - Investigational Site Number 484019, Mexico City
  - Investigational Site Number 484027, México
  - Investigational Site Number 484013, Monterrey
  - Investigational Site Number 484018, Monterrey
  - Investigational Site Number 484011, Monterrey
  - Investigational Site Number 484007, Monterrey
  - Investigational Site Number 484017, Morelia
  - Investigational Site Number 484012, Oaxaca City
  - Investigational Site Number 484014, Querétaro
  - Investigational Site Number 484009, San Luis Potosí City
  - Investigational Site Number 484002, Tijuana
  - Investigational Site Number 484020, Toluca
- Netherlands (32):
  - Investigational Site Number 528006, Alkmaar
  - Investigational Site Number 528022, Amsterdam
  - Investigational Site Number 528026, Amsterdam
  - Investigational Site Number 528021, Apeldoorn
  - Investigational Site Number 528029, Arnhem
  - Investigational Site Number 528004, Breda
  - Investigational Site Number 528002, Delft
  - Investigational Site Number 528007, Eindhoven
  - Investigational Site Number 528032, Goes
  - Investigational Site Number 528012, Gouda
  - Investigational Site Number 528001, Groningen
  - Investigational Site Number 528025, Haarlem
  - Investigational Site Number 528023, Hardenberg
  - Investigational Site Number 528024, Heerenveen
  - Investigational Site Number 528016, Hoorn
  - Investigational Site Number 528019, Leeuwarden
  - Investigational Site Number 528008, Leiden
  - Investigational Site Number 528017, Meppel
  - Investigational Site Number 528030, Nieuwegein
  - Investigational Site Number 528011, Nijmegen
  - Investigational Site Number 528015, Purmerend
  - Investigational Site Number 528018, Roosendaal
  - Investigational Site Number 528014, Rotterdam
  - Investigational Site Number 528027, Rotterdam
  - Investigational Site Number 528005, Sneek
  - Investigational Site Number 528034, Tiel
  - Investigational Site Number 528013, Tilburg
  - Investigational Site Number 528028, Uden
  - Investigational Site Number 528009, Venlo
  - Investigational Site Number 528033, Zaandam
  - Investigational Site Number 528031, Zutphen
  - Investigational Site Number 528020, Zwolle
- New Zealand (12):
  - Investigational Site Number 554010, Auckland
  - Investigational Site Number 554001, Christchurch
  - Investigational Site Number 554006, Dunedin
  - Investigational Site Number 554004, Hamilton
  - Investigational Site Number 554011, Lower Hutt
  - Investigational Site Number 554005, Nelson
  - Investigational Site Number 554007, New Plymouth
  - Investigational Site Number 554002, Otahuhu
  - Investigational Site Number 554008, Palmerston North
  - Investigational Site Number 554012, Rotorua
  - Investigational Site Number 554009, Takapuna
  - Investigational Site Number 554003, Wellington
- North Macedonia (5):
  - Investigational Site Number 807005, Bitola
  - Investigational Site Number 807004, Shtip
  - Investigational Site Number 807002, Skopje
  - Investigational Site Number 807001, Skopje
  - Investigational Site Number 807003, Tetovo
- Norway (9):
  - Investigational Site Number 578004, Arendal
  - Investigational Site Number 578013, Bergen
  - Investigational Site Number 578009, Hamar
  - Investigational Site Number 578006, Kongsvinger
  - Investigational Site Number 578003, Oslo
  - Investigational Site Number 578005, Oslo
  - Investigational Site Number 578012, Stavanger
  - Investigational Site Number 578002, Svelvik
  - Investigational Site Number 578011, Tynset
- Peru (20):
  - Investigational Site Number 604018, Arequipa
  - Investigational Site Number 604004, Callao
  - Investigational Site Number 604025, Callao
  - Investigational Site Number 604022, Cuzco
  - Investigational Site Number 604013, Ica
  - Investigational Site Number 604010, Lima
  - Investigational Site Number 604008, Lima
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604015, Lima
  - Investigational Site Number 604016, Lima
  - Investigational Site Number 604017, Lima
  - Investigational Site Number 604019, Lima
  - Investigational Site Number 604003, Lima
  - Investigational Site Number 604024, Lima
  - Investigational Site Number 604012, Lima
  - Investigational Site Number 604020, Piura
  - Investigational Site Number 604023, Trujillo
- Philippines (13):
  - Investigational Site Number 608012, Cavite
  - Investigational Site Number 608003, Cebu City
  - Investigational Site Number 608013, Cebu City
  - Investigational Site Number 608010, Davao City
  - Investigational Site Number 608011, Davao City
  - Investigational Site Number 608006, Iloilo City
  - Investigational Site Number 608002, Makati City
  - Investigational Site Number 608004, Manila
  - Investigational Site Number 608014, Manila
  - Investigational Site Number 608005, Quezon
  - Investigational Site Number 608001, Quezon City
  - Investigational Site Number 608009, Quezon City
  - Investigational Site Number 608008, San Juan City
- Poland (36):
  - Investigational Site Number 616026, Bydgoszcz
  - Investigational Site Number 616029, Bydgoszcz
  - Investigational Site Number 616010, Chrzanów
  - Investigational Site Number 616036, Czeladź
  - Investigational Site Number 616034, Gdansk
  - Investigational Site Number 616015, Gdansk
  - Investigational Site Number 616035, Gdynia
  - Investigational Site Number 616005, Gdynia
  - Investigational Site Number 616033, Gdynia
  - Investigational Site Number 616037, Grodzisk Mazowiecki
  - Investigational Site Number 616030, Jelenia Góra
  - Investigational Site Number 616031, Krakow
  - Investigational Site Number 616002, Krakow
  - Investigational Site Number 616017, Legnica
  - Investigational Site Number 616019, Lodz
  - Investigational Site Number 616016, Lubin
  - Investigational Site Number 616039, Olsztyn
  - Investigational Site Number 616021, Oława
  - Investigational Site Number 616011, Poznan
  - Investigational Site Number 616018, Puławy
  - Investigational Site Number 616003, Płock
  - Investigational Site Number 616006, Skierniewice
  - Investigational Site Number 616027, Sobótka
  - Investigational Site Number 616007, Sokółka
  - Investigational Site Number 616024, Szczecin
  - Investigational Site Number 616022, Świdnik
  - Investigational Site Number 616004, Torun
  - Investigational Site Number 616013, Torun
  - Investigational Site Number 616025, Torun
  - Investigational Site Number 616032, W?Grów
  - Investigational Site Number 616040, Warsaw
  - Investigational Site Number 616020, Warsaw
  - Investigational Site Number 616038, Warsaw
  - Investigational Site Number 616008, Warsaw
  - Investigational Site Number 616041, Wroclaw
  - Investigational Site Number 616012, Łęczna
- Portugal (9):
  - Investigational Site Number 620004, Almada
  - Investigational Site Number 620005, Aveiro
  - Investigational Site Number 620011, Coimbra
  - Investigational Site Number 620008, Coimbra
  - Investigational Site Number 620001, Leiria
  - Investigational Site Number 620003, Ponta Delgada
  - Investigational Site Number 620002, Setúbal
  - Investigational Site Number 620010, Vila Franca de Xira
  - Investigational Site Number 620006, Vila Nova Gaia
- Romania (17):
  - Investigational Site Number 642001, Brăila
  - Investigational Site Number 642003, Bucharest
  - Investigational Site Number 642012, Bucharest
  - Investigational Site Number 642021, Bucharest
  - Investigational Site Number 642007, Bucharest
  - Investigational Site Number 642008, Bucharest
  - Investigational Site Number 642005, Buzău
  - Investigational Site Number 642013, Codlea
  - Investigational Site Number 642004, Constanța
  - Investigational Site Number 642002, Craiova
  - Investigational Site Number 642016, Craiova
  - Investigational Site Number 642010, Focşani
  - Investigational Site Number 642017, Iași
  - Investigational Site Number 642006, Târgovişte
  - Investigational Site Number 642019, Târgu Mureş
  - Investigational Site Number 642015, Târgu Mureş
  - Investigational Site Number 642018, Timișoara
- Russia (43):
  - Investigational Site Number 643027, Barnaul
  - Investigational Site Number 643037, Kazan'
  - Investigational Site Number 643013, Kemerovo
  - Investigational Site Number 643020, Krasnodar
  - Investigational Site Number 643053, Krasnodar
  - Investigational Site Number 643033, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643011, Moscow
  - Investigational Site Number 643029, Moscow
  - Investigational Site Number 643028, Moscow
  - Investigational Site Number 643004, Moscow
  - Investigational Site Number 643016, Moscow
  - Investigational Site Number 643023, Moscow
  - Investigational Site Number 643044, Moscow
  - Investigational Site Number 643022, Moscow
  - Investigational Site Number 643031, Moscow
  - Investigational Site Number 643043, Nizhny Novgorod
  - Investigational Site Number 643034, Novosibirsk
  - Investigational Site Number 643052, Novosibirsk
  - Investigational Site Number 643050, Novosibirsk
  - Investigational Site Number 643035, Omsk
  - Investigational Site Number 643039, Perm
  - Investigational Site Number 643008, Rostov-on-Don
  - Investigational Site Number 643017, Ryazan
  - Investigational Site Number 643006, Saint Petersburg
  - Investigational Site Number 643015, Saint Petersburg
  - Investigational Site Number 643051, Saint Petersburg
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643030, Saint Petersburg
  - Investigational Site Number 643010, Saint Petersburg
  - Investigational Site Number 643042, Saint Petersburg
  - Investigational Site Number 643007, Saint Petersburg
  - Investigational Site Number 643040, Saint Petersburg
  - Investigational Site Number 643054, Saint Petersburg
  - Investigational Site Number 643012, Saratov
  - Investigational Site Number 643021, Saratov
  - Investigational Site Number 643003, Saratov
  - Investigational Site Number 643014, Saratov
  - Investigational Site Number 643049, Tomsk
  - Investigational Site Number 643019, Tyumen
  - Investigational Site Number 643025, Tyumen
  - Investigational Site Number 643045, Voronezh
  - Investigational Site Number 643009, Yaroslavl
- Serbia (18):
  - Investigational Site Number 688003, Belgrade
  - Investigational Site Number 688005, Belgrade
  - Investigational Site Number 688006, Belgrade
  - Investigational Site Number 688007, Belgrade
  - Investigational Site Number 688008, Belgrade
  - Investigational Site Number 688010, Belgrade
  - Investigational Site Number 688011, Belgrade
  - Investigational Site Number 688013, Belgrade
  - Investigational Site Number 688015, Belgrade
  - Investigational Site Number 688002, Belgrade
  - Investigational Site Number 688009, Kamenitz
  - Investigational Site Number 688012, Kragujevac
  - Investigational Site Number 688016, Leskovac
  - Investigational Site Number 688004, Niš
  - Investigational Site Number 688001, Niška Banja
  - Investigational Site Number 688018, Pančevo
  - Investigational Site Number 688017, Sremska Mitrovica
  - Investigational Site Number 688014, Valjevo
- Singapore (3):
  - Investigational Site Number 702002, Singapore
  - Investigational Site Number 702003, Singapore
  - Investigational Site Number 702001, Singapore
- Slovakia (19):
  - Investigational Site Number 703001, Bardejov
  - Investigational Site Number 703008, Bratislava
  - Investigational Site Number 703020, Bratislava
  - Investigational Site Number 703014, Bratislava
  - Investigational Site Number 703013, Bratislava
  - Investigational Site Number 703023, Dolný Kubín
  - Investigational Site Number 703002, Košice
  - Investigational Site Number 703009, Košice
  - Investigational Site Number 703016, Košice
  - Investigational Site Number 703019, Košice
  - Investigational Site Number 703007, Košice
  - Investigational Site Number 703012, Kráľovský Chlmec
  - Investigational Site Number 703006, Lučenec
  - Investigational Site Number 703010, Lučenec
  - Investigational Site Number 703003, Nitra
  - Investigational Site Number 703004, Prešov
  - Investigational Site Number 703018, Svidník
  - Investigational Site Number 703022, Trebišov
  - Investigational Site Number 703005, Žilina
- Slovenia (5):
  - Investigational Site Number 705001, Celje
  - Investigational Site Number 705004, Izola
  - Investigational Site Number 705002, Jesenice
  - Investigational Site Number 705005, Ljubljana
  - Investigational Site Number 705006, Ljubljana
- South Africa (21):
  - Investigational Site Number 710017, Alberton
  - Investigational Site Number 710007, Bellville
  - Investigational Site Number 710015, Bloemfontein
  - Investigational Site Number 710009, Cape Town
  - Investigational Site Number 710010, Cape Town
  - Investigational Site Number 710005, Chatsworth
  - Investigational Site Number 710006, Durban
  - Investigational Site Number 710004, Durban
  - Investigational Site Number 710002, Durban
  - Investigational Site Number 710012, Johannesburg
  - Investigational Site Number 710014, Johannesburg
  - Investigational Site Number 710019, Kempton Park
  - Investigational Site Number 710011, Kimberley
  - Investigational Site Number 710021, Kuils River
  - Investigational Site Number 710018, Parow
  - Investigational Site Number 710008, Pretoria
  - Investigational Site Number 710016, Pretoria
  - Investigational Site Number 710020, Stellenbosch
  - Investigational Site Number 710013, Tongaat
  - Investigational Site Number 710022, Western Cape
  - Investigational Site Number 710003, Worcester
- South Korea (13):
  - Investigational Site Number 410013, Busan
  - Investigational Site Number 410003, Busan
  - Investigational Site Number 410002, Daegu
  - Investigational Site Number 410012, Goyang-si
  - Investigational Site Number 410001, Gwangju
  - Investigational Site Number 410008, Seongnam
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410007, Seoul
  - Investigational Site Number 410010, Seoul
  - Investigational Site Number 410011, Seoul
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410009, Suwon
  - Investigational Site Number 410005, Wŏnju
- Spain (40):
  - Investigational Site Number 724010, Alcalá de Henares
  - Investigational Site Number 724007, Almería
  - Investigational Site Number 724037, Barcelona
  - Investigational Site Number 724041, Barcelona
  - Investigational Site Number 724038, Barcelona
  - Investigational Site Number 724008, Barcelona
  - Investigational Site Number 724039, Cáceres
  - Investigational Site Number 724042, Córdoba
  - Investigational Site Number 724027, Fuenlabrada
  - Investigational Site Number 724002, Girona
  - Investigational Site Number 724013, Granada
  - Investigational Site Number 724032, Guadalajara
  - Investigational Site Number 724003, Huelva
  - Investigational Site Number 724025, L'Hospitalet de Llobregat
  - Investigational Site Number 724021, León
  - Investigational Site Number 724026, Lleida
  - Investigational Site Number 724006, Lugo
  - Investigational Site Number 724030, Madrid
  - Investigational Site Number 724020, Madrid
  - Investigational Site Number 724015, Madrid
  - Investigational Site Number 724031, Madrid
  - Investigational Site Number 724033, Madrid
  - Investigational Site Number 724017, Madrid
  - Investigational Site Number 724035, Majadahonda
  - Investigational Site Number 724016, Málaga
  - Investigational Site Number 724043, Málaga
  - Investigational Site Number 724036, Murcia
  - Investigational Site Number 724001, Oviedo
  - Investigational Site Number 724022, Sabadell
  - Investigational Site Number 724029, San Sebastián de los Reyes
  - Investigational Site Number 724028, Santander
  - Investigational Site Number 724034, Santiago de Compostela
  - Investigational Site Number 724014, Seville
  - Investigational Site Number 724024, Tarragona
  - Investigational Site Number 724019, Valencia
  - Investigational Site Number 724009, Valencia
  - Investigational Site Number 724011, Valencia
  - Investigational Site Number 724023, Valladolid
  - Investigational Site Number 724005, Vigo
  - Investigational Site Number 724040, Zaragoza
- Sri Lanka (10):
  - Investigational Site Number 144002, Colombo
  - Investigational Site Number 144003, Colombo
  - Investigational Site Number 144004, Colombo
  - Investigational Site Number 144010, Colombo
  - Investigational Site Number 144005, Colombo
  - Investigational Site Number 144006, Colombo
  - Investigational Site Number 144001, Colombo
  - Investigational Site Number 144008, Kandy
  - Investigational Site Number 144009, Kurunegala
  - Investigational Site Number 144007, Ragama
- Sweden (13):
  - Investigational Site Number 752001, Falun
  - Investigational Site Number 752016, Gothenburg
  - Investigational Site Number 752011, Halmstad
  - Investigational Site Number 752006, Karlshamn
  - Investigational Site Number 752008, Karlskrona
  - Investigational Site Number 752013, Köping
  - Investigational Site Number 752004, Kristianstad
  - Investigational Site Number 752015, Malmo
  - Investigational Site Number 752012, Mölndal
  - Investigational Site Number 752009, Stockholm
  - Investigational Site Number 752002, Stockholm
  - Investigational Site Number 752014, Sundsvall
  - Investigational Site Number 752007, Uppsala
- Switzerland (4):
  - Investigational Site Number 756005, Basel
  - Investigational Site Number 756003, Geneva
  - Investigational Site Number 756004, Lugano
  - Investigational Site Number 756002, Zurich
- Taiwan (13):
  - Investigational Site Number 158003, Changhua
  - Investigational Site Number 158008, Division of Cardiology
  - Investigational Site Number 158014, Hsinchu
  - Investigational Site Number 158013, Kaohsiung City
  - Investigational Site Number 158004, Taichung
  - Investigational Site Number 158009, Tainan
  - Investigational Site Number 158011, Tainan
  - Investigational Site Number 158005, Taipei
  - Investigational Site Number 158001, Taipei
  - Investigational Site Number 158010, Taipei
  - Investigational Site Number 158007, Taipei
  - Investigational Site Number 158012, Taoyuan Hsien
  - Investigational Site Number 158002, Yunlin
- Thailand (11):
  - Investigational Site Number 764001, Bangkok
  - Investigational Site Number 764011, Bangkok
  - Investigational Site Number 764007, Bangkok
  - Investigational Site Number 764012, Bangkok
  - Investigational Site Number 764009, Bangkok Noi
  - Investigational Site Number 764005, Hat Yai
  - Investigational Site Number 764008, Klong Luang
  - Investigational Site Number 764002, Moung
  - Investigational Site Number 764003, Muang
  - Investigational Site Number 764010, Nonthaburi
  - Investigational Site Number 764006, Pratumwan
- Turkey (Türkiye) (12):
  - Investigational Site Number 792007, Adana
  - Investigational Site Number 792009, Ankara
  - Investigational Site Number 792006, Bursa
  - Investigational Site Number 792016, Eskişehir
  - Investigational Site Number 792014, Istanbul
  - Investigational Site Number 792005, Istanbul
  - Investigational Site Number 792011, Istanbul
  - Investigational Site Number 792013, Istanbul
  - Investigational Site Number 792004, Izmir
  - Investigational Site Number 792003, Izmir
  - Investigational Site Number 792015, Kocaeli
  - Investigational Site Number 792010, Mersin
- Ukraine (32):
  - Investigational Site Number 804015, Chernivtsi
  - Investigational Site Number 804018, Dnipropetrovsk
  - Investigational Site Number 804027, Donetsk
  - Investigational Site Number 804012, Donetsk
  - Investigational Site Number 804010, Ivano-Frankivsk
  - Investigational Site Number 804006, Kharkiv
  - Investigational Site Number 804003, Kharkiv
  - Investigational Site Number 804009, Kharkiv
  - Investigational Site Number 804020, Khmelnytskyi
  - Investigational Site Number 804001, Kiev
  - Investigational Site Number 804002, Kiev
  - Investigational Site Number 804011, Kyiv
  - Investigational Site Number 804014, Kyiv
  - Investigational Site Number 804025, Kyiv
  - Investigational Site Number 804034, Kyiv
  - Investigational Site Number 804036, Kyiv
  - Investigational Site Number 804016, Kyiv
  - Investigational Site Number 804030, Kyiv
  - Investigational Site Number 804028, Lutsk
  - Investigational Site Number 804033, Lviv
  - Investigational Site Number 804031, Lviv
  - Investigational Site Number 804029, Mykolaiv
  - Investigational Site Number 804004, Odesa
  - Investigational Site Number 804013, Odesa
  - Investigational Site Number 804017, Simferopol
  - Investigational Site Number 804035, Sumy
  - Investigational Site Number 804007, Uzhhorod
  - Investigational Site Number 804005, Vinnitsya
  - Investigational Site Number 804008, Vinnytsia
  - Investigational Site Number 804026, Zaporizhia
  - Investigational Site Number 804024, Zhytomyr
  - Investigational Site Number 804032, Zhytomyr
- United Kingdom (35):
  - Investigational Site Number 826018, Basildon
  - Investigational Site Number 826015, Birmingham
  - Investigational Site Number 826030, Birmingham
  - Investigational Site Number 826038, Bournemouth
  - Investigational Site Number 826025, Bradford
  - Investigational Site Number 826027, Burton-on-Trent
  - Investigational Site Number 826017, Cardiff
  - Investigational Site Number 826010, Chertsey
  - Investigational Site Number 826012, Chesterfield
  - Investigational Site Number 826039, Chichester
  - Investigational Site Number 826024, Cumbria
  - Investigational Site Number 826041, Dudley
  - Investigational Site Number 826021, Harrow
  - Investigational Site Number 826026, High Wycombe
  - Investigational Site Number 826028, Hull
  - Investigational Site Number 826034, London
  - Investigational Site Number 826004, Manchester
  - Investigational Site Number 826011, Newcastle upon Tyne
  - Investigational Site Number 826036, Northampton
  - Investigational Site Number 826019, Peterborough
  - Investigational Site Number 826020, Plymouth
  - Investigational Site Number 826040, Portadown
  - Investigational Site Number 826016, Portsmouth
  - Investigational Site Number 826014, Redhill
  - Investigational Site Number 826007, Rhyl
  - Investigational Site Number 826001, Romford
  - Investigational Site Number 826009, Rotherham
  - Investigational Site Number 826002, Sheffield
  - Investigational Site Number 826032, South Shields
  - Investigational Site Number 826013, St Leonards
  - Investigational Site Number 826005, Stoke-on-Trent
  - Investigational Site Number 826031, Sunderland
  - Investigational Site Number 826022, Truro
  - Investigational Site Number 826035, Wigan
  - Investigational Site Number 826003, Worcester

REFERENCES:
- [Derived] Tsimikas S, Szarek M, Cobbaert CM, Romijn F, Jukema JW, Bhatt DL, Bittner VA, Diaz R, Fazio S, Garon G, Yuan C, Gong XM, Goodman SG, White HD, Witztum JL, Steg PG, Schwartz GG; ODYSSEY OUTCOMES Investigators. Oxidized Phospholipids, Lipoprotein(a), and Cardiovascular Outcomes After Acute Coronary Syndrome. Circulation. 2025 Dec 16;152(24):1666-1678. doi: 10.1161/CIRCULATIONAHA.125.073855. Epub 2025 Dec 1. PMID 41321238
- [Derived] Reijnders E, Bossuyt PM, Jukema JW, Ruhaak LR, Romijn FPHTM, Szarek M, Trompet S, Bhatt DL, Bittner VA, Diaz R, Fazio S, Stevanovic I, Goodman SG, Harrington RA, White HD, Steg PG, Schwartz GG, Cobbaert CM. Multiplex Apolipoprotein Panel Improves Cardiovascular Event Prediction and Cardiovascular Outcome by Identifying Patients Who Benefit From Targeted PCSK9 Inhibitor Therapy. Arterioscler Thromb Vasc Biol. 2025 Nov;45(11):2111-2123. doi: 10.1161/ATVBAHA.124.322336. Epub 2025 Sep 25. PMID 40995631
- [Derived] Geba GP, Mohammadi KA, Damask A, Paulding C, Lotta LA, Hindy G, Pordy R, Manvelian G, Shapiro MD, Bittner VA, Bhatt DL, Szarek M, Schwartz GG, Steg PG, Fazio S. Effect of PCSK9 Inhibition With Alirocumab in Patients With Probable Familial Hypercholesterolemia or Type III Hyperlipoproteinemia: Results From the ODYSSEY OUTCOMES Trial. J Am Heart Assoc. 2025 Sep 2;14(17):e041190. doi: 10.1161/JAHA.124.041190. Epub 2025 Aug 22. PMID 40847481
- [Derived] Steg PG, Szarek M, Jukema JW, Bhatt DL, Bittner VA, Diaz R, Fazio S, Garon G, Goodman SG, Harrington RA, White HD, Zeiher AM, Schwartz GG; ODYSSEY OUTCOMES Investigators. Relation of Low-Density Lipoprotein Cholesterol, High-Sensitivity C-Reactive Protein, and Lipoprotein(a) Each to Future Cardiovascular Events and Death After Acute Coronary Syndrome on High-Intensity Statin Therapy: An Analysis of the Placebo Arm of ODYSSEY OUTCOMES. Circulation. 2025 Apr 8;151(14):1047-1050. doi: 10.1161/CIRCULATIONAHA.124.071269. Epub 2025 Apr 7. No abstract available. PMID 40193536
- [Derived] Geba GP, Chen R, Talapatra K, Brackin T, Mohammadi KA, Pordy R, Manvelian G, Maron DJ, Schwartz GG, Szarek M, Steg PG, Fazio S. Alirocumab and chest pain after acute coronary syndrome: An analysis of ODYSSEY OUTCOMES. Am J Prev Cardiol. 2024 Nov 26;20:100900. doi: 10.1016/j.ajpc.2024.100900. eCollection 2024 Dec. PMID 39687787
- [Derived] Reijnders E, Romijn FPHTM, Arslan F, Georges JJJ, Pieterse MM, Schipper ER, Didden-Buitendijk S, Martherus-Bultman MC, Smit NPM, Diederiks NM, Treep MM, Jukema JW, Cobbaert CM, Ruhaak LR. Quality Assurance for Multiplex Quantitative Clinical Chemistry Proteomics in Large Clinical Trials. J Appl Lab Med. 2024 Nov 4;9(6):949-963. doi: 10.1093/jalm/jfae092. PMID 39239905
- [Derived] Zahger D, Schwartz GG, Du W, Szarek M, Bhatt DL, Bittner VA, Budaj AJ, Diaz R, Goodman SG, Jukema JW, Kiss RG, Harrington RA, Moriarty PM, Scemama M, Manvelian G, Pordy R, White HD, Zeiher AM, Fazio S, Geba GP, Steg PG; ODYSSEY OUTCOMES Investigators. Triglyceride Levels, Alirocumab Treatment, and Cardiovascular Outcomes After an Acute Coronary Syndrome. J Am Coll Cardiol. 2024 Sep 10;84(11):994-1006. doi: 10.1016/j.jacc.2024.06.035. PMID 39232634
- [Derived] Lawler PR, Manvelian G, Coppi A, Damask A, Cantor MN, Ferreira MAR, Paulding C, Banerjee N, Li D, Jorgensen S, Attre R, Carey DJ, Krebs K, Milani L, Hveem K, Damas JK, Solligard E, Stender S, Tybjaerg-Hansen A, Nordestgaard BG, Hernandez-Beeftink T, Rogne T, Flores C, Villar J, Walley KR, Liu VX, Fohner AE, Lotta LA, Kyratsous CA, Sleeman MW, Scemama M, DelGizzi R, Pordy R, Horowitz JE, Baras A, Martin GS, Steg PG, Schwartz GG, Szarek M, Goodman SG. Pharmacologic and Genetic Downregulation of Proprotein Convertase Subtilisin/Kexin Type 9 and Survival From Sepsis. Crit Care Explor. 2023 Nov 8;5(11):e0997. doi: 10.1097/CCE.0000000000000997. eCollection 2023 Nov. PMID 37954898
- [Derived] Goodman SG, Steg PG, Poulouin Y, Bhatt DL, Bittner VA, Diaz R, Garon G, Harrington RA, Jukema JW, Manvelian G, Stipek W, Szarek M, White HD, Schwartz GG; ODYSSEY OUTCOMES Investigators. Long-Term Efficacy, Safety, and Tolerability of Alirocumab in 8242 Patients Eligible for 3 to 5 Years of Placebo-Controlled Observation in the ODYSSEY OUTCOMES Trial. J Am Heart Assoc. 2023 Sep 19;12(18):e029216. doi: 10.1161/JAHA.122.029216. Epub 2023 Sep 13. No abstract available. PMID 37702079
- [Derived] Szarek M, Reijnders E, Jukema JW, Bhatt DL, Bittner VA, Diaz R, Fazio S, Garon G, Goodman SG, Harrington RA, Ruhaak LR, Schwertfeger M, Tsimikas S, White HD, Steg PG, Cobbaert C, Schwartz GG; ODYSSEY OUTCOMES Investigators. Relating Lipoprotein(a) Concentrations to Cardiovascular Event Risk After Acute Coronary Syndrome: A Comparison of 3 Tests. Circulation. 2024 Jan 16;149(3):192-203. doi: 10.1161/CIRCULATIONAHA.123.066398. Epub 2023 Aug 26. PMID 37632469
- [Derived] Suc G, Schwartz GG, Goodman SG, Jukema JW, Manvelian G, Poulouin Y, Pordy R, Scemama M, Szarek M, Steg PG; ODYSSEY OUTCOMES Investigators. Effect of alirocumab on cataracts in patients with acute coronary syndromes. BMC Ophthalmol. 2023 Jun 16;23(1):279. doi: 10.1186/s12886-023-03012-1. PMID 37328736
- [Derived] Schwartz GG, Szarek M, Bhatt DL, Bittner VA, Bujas-Bobanovic M, Diaz R, Fazio S, Fras Z, Goodman SG, Harrington RA, Jukema JW, Manvelian G, Pordy R, Ray KK, Scemama M, White HD, Steg PG; ODYSSEY OUTCOMES Investigators. Transiently achieved very low LDL-cholesterol levels by statin and alirocumab after acute coronary syndrome are associated with cardiovascular risk reduction: the ODYSSEY OUTCOMES trial. Eur Heart J. 2023 Mar 5;44(16):1408-17. doi: 10.1093/eurheartj/ehad144. Online ahead of print. PMID 36879424
- [Derived] Hagstrom E, Steg PG, Szarek M, Bhatt DL, Bittner VA, Danchin N, Diaz R, Goodman SG, Harrington RA, Jukema JW, Liberopoulos E, Marx N, McGinniss J, Manvelian G, Pordy R, Scemama M, White HD, Zeiher AM, Schwartz GG; ODYSSEY OUTCOMES Investigators. Apolipoprotein B, Residual Cardiovascular Risk After Acute Coronary Syndrome, and Effects of Alirocumab. Circulation. 2022 Aug 30;146(9):657-672. doi: 10.1161/CIRCULATIONAHA.121.057807. Epub 2022 Jun 30. PMID 35770629
- [Derived] Landmesser U, McGinniss J, Steg PG, Bhatt DL, Bittner VA, Diaz R, Dilic M, Goodman SG, Jukema JW, Loy M, Pecin I, Pordy R, Poulsen SH, Szarek M, White HD, Schwartz GG; ODYSSEY OUTCOMES Investigators. Achievement of ESC/EAS LDL-C treatment goals after an acute coronary syndrome with statin and alirocumab. Eur J Prev Cardiol. 2022 Oct 20;29(14):1842-1851. doi: 10.1093/eurjpc/zwac107. PMID 35708715
- [Derived] Chiang CE, Schwartz GG, Elbez Y, Szarek M, Bhatt DL, Bittner VA, Diaz R, Erglis A, Goodman SG, Hagstrom E, Jukema JW, Liberopoulos E, Loy M, Pordy R, White HD, Simon T, Steg PG; ODYSSEY OUTCOMES Investigators. Alirocumab and Cardiovascular Outcomes in Patients With Previous Myocardial Infarction: Prespecified Subanalysis From ODYSSEY OUTCOMES. Can J Cardiol. 2022 Oct;38(10):1542-1549. doi: 10.1016/j.cjca.2022.05.021. Epub 2022 May 27. PMID 35644332
- [Derived] Ostadal P, Steg PG, Poulouin Y, Bhatt DL, Bittner VA, Chua T, Diaz R, Goodman SG, Huo Y, Jukema JW, Karpov Y, Pordy R, Scemama M, Szarek M, White HD, Schwartz GG; ODYSSEY OUTCOMES Investigators. Metabolic risk factors and effect of alirocumab on cardiovascular events after acute coronary syndrome: a post-hoc analysis of the ODYSSEY OUTCOMES randomised controlled trial. Lancet Diabetes Endocrinol. 2022 May;10(5):330-340. doi: 10.1016/S2213-8587(22)00043-2. Epub 2022 Apr 1. PMID 35378068
- [Derived] Lopes RD, Guimaraes PO, Schwartz GG, Bhatt DL, Bittner VA, Budaj A, Dalby AJ, Diaz R, Goodman SG, Harrington RA, Jukema JW, Kiss RG, Loy M, Pordy R, Poulouin Y, Szarek M, White HD, Steg PG; ODYSSEY OUTCOMES Investigators. Effect of Alirocumab on Incidence of Atrial Fibrillation After Acute Coronary Syndromes: Insights from the ODYSSEY OUTCOMES Trial. Am J Med. 2022 Jul;135(7):915-918. doi: 10.1016/j.amjmed.2022.02.016. Epub 2022 Mar 14. PMID 35296402
- [Derived] Schwartz GG, Szarek M, Bittner VA, Diaz R, Goodman SG, Jukema JW, Landmesser U, Lopez-Jaramillo P, Manvelian G, Pordy R, Scemama M, Sinnaeve PR, White HD, Gabriel Steg P; ODYSSEY Outcomes Committees and Investigators. Lipoprotein(a) and Benefit of PCSK9 Inhibition in Patients With Nominally Controlled LDL Cholesterol. J Am Coll Cardiol. 2021 Aug 3;78(5):421-433. doi: 10.1016/j.jacc.2021.04.102. PMID 34325831
- [Derived] Diaz R, Li QH, Bhatt DL, Bittner VA, Baccara-Dinet MT, Goodman SG, Jukema JW, Kimura T, Parkhomenko A, Pordy R, Reiner Z, Roe MT, Szarek M, Tse HF, White HD, Zahger D, Zeiher AM, Schwartz GG, Steg PG; ODYSSEY OUTCOMES Committees and Investigators. Intensity of statin treatment after acute coronary syndrome, residual risk, and its modification by alirocumab: insights from the ODYSSEY OUTCOMES trial. Eur J Prev Cardiol. 2021 Mar 23;28(1):33-43. doi: 10.1177/2047487320941987. Epub 2020 Jul 27. PMID 33755145
- [Derived] Schwartz GG, Szarek M, Bittner VA, Bhatt DL, Diaz R, Goodman SG, Jukema JW, Loy M, Manvelian G, Pordy R, White HD, Steg PG; ODYSSEY OUTCOMES Committees and Investigators. Relation of Lipoprotein(a) Levels to Incident Type 2 Diabetes and Modification by Alirocumab Treatment. Diabetes Care. 2021 May;44(5):1219-1227. doi: 10.2337/dc20-2842. Epub 2021 Mar 15. PMID 33722880
- [Derived] Schwartz GG, Gabriel Steg P, Bhatt DL, Bittner VA, Diaz R, Goodman SG, Jukema JW, Kim YU, Li QH, Manvelian G, Pordy R, Sourdille T, White HD, Szarek M; ODYSSEY OUTCOMES Committees and Investigators. Clinical Efficacy and Safety of Alirocumab After Acute Coronary Syndrome According to Achieved Level of Low-Density Lipoprotein Cholesterol: A Propensity Score-Matched Analysis of the ODYSSEY OUTCOMES Trial. Circulation. 2021 Mar 16;143(11):1109-1122. doi: 10.1161/CIRCULATIONAHA.120.049447. Epub 2021 Jan 13. PMID 33438437
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Szarek M, Bittner VA, Aylward P, Baccara-Dinet M, Bhatt DL, Diaz R, Fras Z, Goodman SG, Halvorsen S, Harrington RA, Jukema JW, Moriarty PM, Pordy R, Ray KK, Sinnaeve P, Tsimikas S, Vogel R, White HD, Zahger D, Zeiher AM, Steg PG, Schwartz GG; ODYSSEY OUTCOMES Investigators. Lipoprotein(a) lowering by alirocumab reduces the total burden of cardiovascular events independent of low-density lipoprotein cholesterol lowering: ODYSSEY OUTCOMES trial. Eur Heart J. 2020 Nov 21;41(44):4245-4255. doi: 10.1093/eurheartj/ehaa649. PMID 33051646
- [Derived] Bhatt DL, Briggs AH, Reed SD, Annemans L, Szarek M, Bittner VA, Diaz R, Goodman SG, Harrington RA, Higuchi K, Joulain F, Jukema JW, Li QH, Mahaffey KW, Sanchez RJ, Roe MT, Lopes RD, White HD, Zeiher AM, Schwartz GG, Gabriel Steg P; ODYSSEY OUTCOMES Investigators. Cost-Effectiveness of Alirocumab in Patients With Acute Coronary Syndromes: The ODYSSEY OUTCOMES Trial. J Am Coll Cardiol. 2020 May 12;75(18):2297-2308. doi: 10.1016/j.jacc.2020.03.029. PMID 32381160
- [Derived] Schwartz GG, Steg PG, Szarek M, Bittner VA, Diaz R, Goodman SG, Kim YU, Jukema JW, Pordy R, Roe MT, White HD, Bhatt DL; ODYSSEY OUTCOMES Committees and Investigators*. Peripheral Artery Disease and Venous Thromboembolic Events After Acute Coronary Syndrome: Role of Lipoprotein(a) and Modification by Alirocumab: Prespecified Analysis of the ODYSSEY OUTCOMES Randomized Clinical Trial. Circulation. 2020 May 19;141(20):1608-1617. doi: 10.1161/CIRCULATIONAHA.120.046524. Epub 2020 Mar 29. PMID 32223446
- [Derived] Bittner VA, Szarek M, Aylward PE, Bhatt DL, Diaz R, Edelberg JM, Fras Z, Goodman SG, Halvorsen S, Hanotin C, Harrington RA, Jukema JW, Loizeau V, Moriarty PM, Moryusef A, Pordy R, Roe MT, Sinnaeve P, Tsimikas S, Vogel R, White HD, Zahger D, Zeiher AM, Steg PG, Schwartz GG; ODYSSEY OUTCOMES Committees and Investigators. Effect of Alirocumab on Lipoprotein(a) and Cardiovascular Risk After Acute Coronary Syndrome. J Am Coll Cardiol. 2020 Jan 21;75(2):133-144. doi: 10.1016/j.jacc.2019.10.057. PMID 31948641
- [Derived] Szarek M, Steg PG, DiCenso D, Bhatt DL, Bittner VA, Budaj A, Diaz R, Goodman SG, Gotcheva N, Jukema JW, Pordy R, Roe MT, Sourdille T, White HD, Xavier D, Zeiher AM, Schwartz GG. Alirocumab Reduces Total Hospitalizations and Increases Days Alive and Out of Hospital in the ODYSSEY OUTCOMES Trial. Circ Cardiovasc Qual Outcomes. 2019 Nov;12(11):e005858. doi: 10.1161/CIRCOUTCOMES.119.005858. Epub 2019 Nov 11. PMID 31707826
- [Derived] Jukema JW, Zijlstra LE, Bhatt DL, Bittner VA, Diaz R, Drexel H, Goodman SG, Kim YU, Pordy R, Reiner Z, Roe MT, Tse HF, Montenegro Valdovinos PC, White HD, Zeiher AM, Szarek M, Schwartz GG, Steg PG; ODYSSEY OUTCOMES Investigators. Effect of Alirocumab on Stroke in ODYSSEY OUTCOMES. Circulation. 2019 Dec 17;140(25):2054-2062. doi: 10.1161/CIRCULATIONAHA.119.043826. Epub 2019 Nov 11. PMID 31707788
- [Derived] Roe MT, Li QH, Bhatt DL, Bittner VA, Diaz R, Goodman SG, Harrington RA, Jukema JW, Lopez-Jaramillo P, Lopes RD, Louie MJ, Moriarty PM, Szarek M, Vogel R, White HD, Zeiher AM, Baccara-Dinet MT, Steg PG, Schwartz GG. Risk Categorization Using New American College of Cardiology/American Heart Association Guidelines for Cholesterol Management and Its Relation to Alirocumab Treatment Following Acute Coronary Syndromes. Circulation. 2019 Nov 5;140(19):1578-1589. doi: 10.1161/CIRCULATIONAHA.119.042551. Epub 2019 Sep 2. PMID 31475572
- [Derived] Goodman SG, Aylward PE, Szarek M, Chumburidze V, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Hanotin C, Harrington RA, Jukema JW, Kedev S, Letierce A, Moryusef A, Pordy R, Ramos Lopez GA, Roe MT, Viigimaa M, White HD, Zeiher AM, Steg PG, Schwartz GG; ODYSSEY OUTCOMES Committees and Investigators. Effects of Alirocumab on Cardiovascular Events After Coronary Bypass Surgery. J Am Coll Cardiol. 2019 Sep 3;74(9):1177-1186. doi: 10.1016/j.jacc.2019.07.015. PMID 31466614
- [Derived] Ray KK, Colhoun HM, Szarek M, Baccara-Dinet M, Bhatt DL, Bittner VA, Budaj AJ, Diaz R, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Loizeau V, Lopes RD, Moryusef A, Murin J, Pordy R, Ristic AD, Roe MT, Tunon J, White HD, Zeiher AM, Schwartz GG, Steg PG; ODYSSEY OUTCOMES Committees and Investigators. Effects of alirocumab on cardiovascular and metabolic outcomes after acute coronary syndrome in patients with or without diabetes: a prespecified analysis of the ODYSSEY OUTCOMES randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Aug;7(8):618-628. doi: 10.1016/S2213-8587(19)30158-5. Epub 2019 Jul 1. PMID 31272931
- [Derived] Steg PG, Szarek M, Bhatt DL, Bittner VA, Bregeault MF, Dalby AJ, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Ostadal P, Parkhomenko A, Pordy R, Roe MT, Tricoci P, Vogel R, White HD, Zeiher AM, Schwartz GG. Effect of Alirocumab on Mortality After Acute Coronary Syndromes. Circulation. 2019 Jul 9;140(2):103-112. doi: 10.1161/CIRCULATIONAHA.118.038840. Epub 2019 May 23. PMID 31117810
- [Derived] Jukema JW, Szarek M, Zijlstra LE, de Silva HA, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Karpov Y, Moryusef A, Pordy R, Prieto JC, Roe MT, White HD, Zeiher AM, Schwartz GG, Steg PG; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab in Patients With Polyvascular Disease and Recent Acute Coronary Syndrome: ODYSSEY OUTCOMES Trial. J Am Coll Cardiol. 2019 Sep 3;74(9):1167-1176. doi: 10.1016/j.jacc.2019.03.013. Epub 2019 Mar 18. PMID 30898609
- [Derived] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Derived] Schwartz GG, Bessac L, Berdan LG, Bhatt DL, Bittner V, Diaz R, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Mahaffey KW, Moryusef A, Pordy R, Roe MT, Rorick T, Sasiela WJ, Shirodaria C, Szarek M, Tamby JF, Tricoci P, White H, Zeiher A, Steg PG. Effect of alirocumab, a monoclonal antibody to PCSK9, on long-term cardiovascular outcomes following acute coronary syndromes: rationale and design of the ODYSSEY outcomes trial. Am Heart J. 2014 Nov;168(5):682-9. doi: 10.1016/j.ahj.2014.07.028. Epub 2014 Aug 7. PMID 25440796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1387 sites in 57 countries. Of these, 1328 active sites randomized at least 1 participant. Overall, 35,437 participants were screened between 11 October 2012 and 17 Jan 2017; of whom 16,513 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to country. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1 ratio (alirocumab: placebo), with permuted-block randomization.
Groups:
- Placebo: Placebo (for alirocumab) SC injection every 2 weeks (Q2W) added to stable Lipid-Modifying Therapy (LMT) for up to 64 months.
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable LMT for up to 64 months. Alirocumab dose up-titrated to 150 mg Q2W from Month 2 when LDL-C levels >=50 mg/dL (1.29 mmol/L) at Month 1; or if up-titration was missed due to unavailability of LDL-C value, it was up-titrated at month 4 based on LDL-C value at Month 2. For participants receiving 150 mg Q2W, alirocumab dose was down-titrated in a blinded manner to 75 mg Q2W if two consecutive values of LDL-C were <25 mg/dL (0.65 mmol/L). For participants receiving 75 mg Q2W, alirocumab dose was switched to placebo in a blinded manner if two consecutive values of LDL-C were <15 mg/dL (0.39 mmol/L).
Period: Overall Study
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Started | 9462 | 9462
Treated | 9443 | 9451
Completed | 7947 | 7378
Not Completed | 1515 | 2084
Not completed — Randomized but not treated | 19 | 11
Not completed — Adverse Event | 347 | 362
Not completed — Two consecutive LDL-C <15 mg/dL | 0 | 730
Not completed — Poor compliance to protocol | 529 | 454
Not completed — Physician Decision | 77 | 62
Not completed — Site terminated by sponsor | 1 | 3
Not completed — Participant moved | 139 | 104
Not completed — Withdrawal by Subject | 118 | 91
Not completed — Related to study drug administration | 96 | 105
Not completed — Lost to Follow-up | 17 | 15
Not completed — Other than specified above | 172 | 147

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Placebo: Placebo (for alirocumab) SC injection Q2W added to stable LMT for up to 64 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Total
Number analyzed (Participants) | 9462 | 9462 | 18924
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.4) | 58.5 (9.3) | 58.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2372 | 2390 | 4762
  Male | 7090 | 7072 | 14162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1555 | 1581 | 3136
  Not Hispanic or Latino | 7721 | 7700 | 15421
  Unknown or Not Reported | 186 | 181 | 367
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Here, 'number analyzed' signifies participants with available for specified measure.
  Participants
    White: number analyzed (Participants) | 9460 | 9461 | 18921
    White | 7524 | 7500 | 15024
    Black or African American: number analyzed (Participants) | 9460 | 9461 | 18921
    Black or African American | 238 | 235 | 473
    Asian: number analyzed (Participants) | 9460 | 9461 | 18921
    Asian | 1247 | 1251 | 2498
    Other: number analyzed (Participants) | 9460 | 9461 | 18921
    Other | 449 | 469 | 918
    Unknown: number analyzed (Participants) | 9460 | 9461 | 18921
    Unknown | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Major Adverse Cardiovascular Event (MACE); Percentage of Observed Participants With Outcome Measure Events During the Study
Description: All MACE positively adjudicated by Clinical Events Committee (CEC) in a blinded fashion, were used in the analysis of the composite cardiovascular (CV) outcome measure comprised of Coronary Heart Disease (CHD) death, non-fatal Myocardial Infarction (MI), fatal and non-fatal ischemic stroke (IS), or unstable angina (UA) requiring hospitalization. Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of MACE over time. Percentage of observed participants with outcome measure events during the study were reported.
Time Frame: From randomization up to 64 months
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 11.1 | 9.5
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Analysis was performed using Cox proportional hazard model and log rank test stratified on geographical region (North America, South America, Western Europe, Eastern Europe, Asia, Rest of the world); Test type: Superiority; p = 0.0003, Log Rank — Threshold for statistical significance at 0.0498 level; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.78 to 0.93]

2. Secondary Outcome: Time to First Occurrence of Any Coronary Heart Disease Event; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: All CHD events positively adjudicated by CEC in a blinded fashion, were used in the analysis of the composite CHD endpoint comprised of any CHD death, non-fatal non-fatal MI, UA requiring hospitalization, or ischemia-driven coronary revascularization procedure. Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any CHD event over time. Percentage of observed participants with outcome measure events during the study were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 14.3 | 12.7
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Analysis was performed using Cox proportional hazard model and log rank test stratified on geographical region(North America,South America,Western Europe,Eastern Europe,Asia, Rest of the world).A hierarchical testing approach was used to control the overall type-I error at 0.0249 one-sided alpha level(0.0498 two-sided).Testing was then performed sequentially in the order endpoints were reported.Hierarchical testing sequence continued only if the previous endpoint was statistically significant; Test type: Superiority; p = 0.0013, Log Rank — Threshold for statistical significance at 0.0498 level; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.81 to 0.95]

3. Secondary Outcome: Time to First Occurrence of Any Major Coronary Heart Disease Event; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: All Major CHD events positively adjudicated by CEC in a blinded fashion, were used in the analysis of the composite CHD endpoint comprised of any CHD death and non-fatal MI. Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any major CHD event over time. Percentage of observed participants with outcome measure events during the study were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 9.5 | 8.4
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Analysis was performed using Cox proportional hazard model and log rank test stratified on geographical region (North America, South America, Western Europe, Eastern Europe, Asia, Rest of the world). Testing was performed according to the hierarchical testing procedure (continued only if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0060, Log Rank — Threshold for statistical significance at 0.0498 level; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.80 to 0.96]

4. Secondary Outcome: Time to First Occurrence of Any Cardiovascular Event; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: All CV events positively adjudicated by CEC in a blinded fashion, were used in the analysis of the composite CV endpoint comprised of any non-fatal CHD event, any CV death and non-fatal IS. Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any CV event over time. Percentage of observed participants with outcome measure events during the study were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 15.6 | 13.7
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Analysis was performed using Cox proportional hazard model and log rank test stratified on geographical region (North America, South America, Western Europe, Eastern Europe, Asia, Rest of the world). Testing according to the hierarchical testing procedure (continued only if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0003, Log Rank — Threshold for statistical significance at 0.0498 level; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.81 to 0.94]

5. Secondary Outcome: Time to First Occurrence of All-Cause Mortality, Non-Fatal Myocardial Infarction, Non-Fatal Ischemic Stroke; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: All-cause mortality, non-fatal MI and non-fatal IS positively adjudicated by CEC in a blinded fashion, were used in the analysis of this endpoint. Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of all-cause mortality, non-fatal MI and non-fatal IS over time. Percentage of observed participants with outcome measure events during the study were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 11.9 | 10.3
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0003, Log Rank — Threshold for statistical significance at 0.0498 level; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.79 to 0.93]

6. Secondary Outcome: Time to Coronary Heart Disease Death; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the CHD death over time. Percentage of observed participants with CHD death (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 2.3 | 2.2
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.3824, Log Rank — Threshold for statistical significance at 0.0498 level; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.76 to 1.11]

7. Secondary Outcome: Time to Cardiovascular Death; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the CV death over time. Percentage of observed participants with CV death (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 2.9 | 2.5

8. Secondary Outcome: Time to All-Cause Death; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the all-cause death over time. Percentage of observed participants with all-cause death (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 4.1 | 3.5

9. Secondary Outcome: Time to First Occurrence of Any Non-Fatal Myocardial Infarction; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any non-fatal MI over time. Percentage of observed participants with any non-fatal MI (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 7.6 | 6.6

10. Secondary Outcome: Time to First Occurrence of Fatal or Any Non-Fatal Ischemic Stroke; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of fatal or any non-fatal IS over time. Percentage of observed participants with fatal or any non-fatal IS (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 1.6 | 1.2

11. Secondary Outcome: Time to First Occurrence of Any Unstable Angina Requiring Hospitalization; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any UA requiring hospitalization over time. Percentage of observed participants with any UA requiring hospitalization (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 0.6 | 0.4

12. Secondary Outcome: Time to First Occurrence of Any Ischemia-Driven Coronary Revascularization Procedure; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any ischemia-driven coronary revascularization procedure over time. Percentage of observed participants with any ischemia-driven coronary revascularization procedure (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 8.8 | 7.7

13. Secondary Outcome: Time to First Occurrence of Any Congestive Heart Failure (CHF) Requiring Hospitalization; Percentage of Observed Participants With Outcome Measure Events During the Study
Description: Kaplan Meier plots of the cumulative incidence rate by treatment groups were used to depict the first occurrence of any CHF requiring hospitalization over time. Percentage of observed participants with any CHF requiring hospitalization (positively adjudicated by CEC in a blinded fashion) were reported.
Time Frame: From randomization up to 64 months
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
percentage of participants | 1.9 | 1.9

14. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Months 4, 12, and 48: ITT Analysis
Description: Adjusted means and standard errors at Month 4, 12 and 48 from multiple imputation approach (to account for missing data) followed by analyses of covariance (ANCOVA) model with the fixed categorical effect of treatment group and the continuous fixed covariate of baseline LDL-C value, including all available post-baseline data from Month 1 up to Month 48 regardless of status on- or off-treatment.
Time Frame: Baseline, Months 4, 12 and 48
Population: ITT Population. Here, 'number analyzed' corresponds to the number of participants with the parameter measured and baseline measure available for each time-point. A multiple approach was used to account for participants with missing data.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9462 | 9462
Percent change
  Month 4: number analyzed (Participants) | 8750 | 8602
  Month 4 | 4.4 (0.3) | -55.8 (0.3)
  Month 12: number analyzed (Participants) | 8397 | 8336
  Month 12 | 8.0 (0.4) | -45.7 (0.4)
  Month 48: number analyzed (Participants) | 790 | 812
  Month 48 | 16.4 (1.8) | -23.5 (1.6)

15. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Months 4, 12, and 48: On-Treatment Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Month 4, 12 and 48 were obtained from a mixed-effect model with repeated measures (MMRM) including available post-baseline on-treatment data from Month 1 up to Month 48 (i.e. up to 21 days after last injection).
Time Frame: Baseline, Months 4, 12 and 48
Population: Randomized and treated population. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 9443 | 9451
Percent change
  Month 4: number analyzed (Participants) | 8647 | 8486
  Month 4 | 4.4 (0.3) | -58.3 (0.3)
  Month 12: number analyzed (Participants) | 8183 | 7727
  Month 12 | 8.2 (0.4) | -52.8 (0.4)
  Month 48: number analyzed (Participants) | 726 | 647
  Month 48 | 14.6 (1.0) | -40.1 (1.0)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form until the end of study (Month 64) regardless of seriousness or relationship to Investigational Medicinal Product (IMP).
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days). Safety population included randomized participants who actually received at least 1 dose or part of a dose of the double-blind IMP injection.
Groups:
- Alirocumab: Alirocumab 75 mg SC injection Q2W added to stable LMT for up to 64 months. Alirocumab dose up-titrated to 150 mg Q2W from Month 2 when LDL-C levels >=50 mg/dL (1.29 mmol/L) at Month 1; or if up-titration was missed due to unavailability of LDL-C value, it was up-titrated at month 4 based on LDL-C value at Month 2. For participants receiving 150 mg Q2W, alirocumab dose was down-titrated in a blinded manner to 75 mg Q2W if two consecutive values of LDL-C were <25 mg/dL (0.65 mmol/L). For participants receiving 75 mg Q2W, alirocumab dose was switched to placebo in a blinded manner if two consecutive values of LDL-C were <15 mg/dL (0.39 mmol/L).
Arm/Group | Placebo | Alirocumab
All-Cause Mortality (participants affected / at risk) | 278/9443 | 238/9451
Serious Adverse Events (participants affected / at risk) | 2350/9443 | 2202/9451
Other Adverse Events (participants affected / at risk) | 2181/9443 | 2203/9451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9443) | Alirocumab (N=9451)
Anaemia (Blood and lymphatic system disorders) | 15 (15) | 11 (11)
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 17 (18) | 14 (15)
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 8 (8) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 2 (2)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 6 (6)
Adams-Stokes Syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 133 (148) | 113 (136)
Angina Unstable (Cardiac disorders) | 8 (8) | 10 (10)
Aortic Valve Disease Mixed (Cardiac disorders) | 2 (2) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1) | 4 (4)
Aortic Valve Sclerosis (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 17 (17) | 7 (7)
Arrhythmia (Cardiac disorders) | 1 (1) | 5 (5)
Arrhythmia Supraventricular (Cardiac disorders) | 2 (2) | 3 (3)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 4 (4) | 2 (2)
Arteriospasm Coronary (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 98 (110) | 82 (103)
Atrial Flutter (Cardiac disorders) | 10 (14) | 14 (16)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 6 (6) | 5 (5)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular Block Second Degree (Cardiac disorders) | 5 (5) | 3 (3)
Bradycardia (Cardiac disorders) | 9 (9) | 8 (8)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Aneurysm (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 9 (10) | 9 (9)
Cardiac Discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 4 (4) | 4 (4)
Cardiac Failure Acute (Cardiac disorders) | 3 (4) | 2 (2)
Cardiac Failure Chronic (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 5 (5) | 4 (4)
Cardiac Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 3 (3) | 4 (4)
Cardiogenic Shock (Cardiac disorders) | 6 (6) | 4 (4)
Cardiomyopathy (Cardiac disorders) | 6 (6) | 1 (1)
Chordae Tendinae Rupture (Cardiac disorders) | 1 (1) | 0 (0)
Conduction Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Coronary Artery Disease (Cardiac disorders) | 20 (20) | 25 (26)
Coronary Artery Dissection (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 3 (3)
Coronary Artery Stenosis (Cardiac disorders) | 3 (3) | 6 (6)
Diastolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac Mass (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 4 (4) | 2 (2)
Ischaemic Cardiomyopathy (Cardiac disorders) | 9 (9) | 9 (9)
Ischaemic Mitral Regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 3 (3) | 2 (2)
Low Cardiac Output Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 7 (7) | 9 (9)
Mitral Valve Prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 4 (4) | 2 (2)
Myocardial Ischaemia (Cardiac disorders) | 13 (13) | 4 (4)
Myocardial Rupture (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nodal Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal Rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 5 (5) | 2 (2)
Papillary Muscle Rupture (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 5 (5) | 3 (3)
Pericardial Haemorrhage (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 6 (6)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal Angina (Cardiac disorders) | 1 (3) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 3 (3) | 1 (1)
Rhythm Idioventricular (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 4 (4)
Sinus Node Dysfunction (Cardiac disorders) | 9 (9) | 13 (13)
Sinus Tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Stress Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 12 (16) | 9 (11)
Systolic Dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tricuspid Valve Disease (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular Extrasystoles (Cardiac disorders) | 5 (5) | 7 (7)
Ventricular Fibrillation (Cardiac disorders) | 17 (17) | 8 (8)
Ventricular Hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 29 (33) | 24 (28)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bicuspid Aortic Valve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Bronchogenic Cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dermoid Cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hereditary Optic Atrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Spinocerebellar Ataxia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thyroglossal Cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Von Hippel-Lindau Disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Acute Vestibular Syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 12 (12) | 9 (9)
Vertigo Labyrinthine (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Adrenal Insufficiency (Endocrine disorders) | 3 (3) | 0 (0)
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1 (1) | 0 (0)
Adrenocorticotropic Hormone Deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Autoimmune Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Basedow's Disease (Endocrine disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 (1) | 1 (1)
Pituitary Cyst (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid Mass (Endocrine disorders) | 1 (1) | 1 (1)
Toxic Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Toxic Nodular Goitre (Endocrine disorders) | 2 (2) | 2 (2)
Amaurosis Fugax (Eye disorders) | 1 (1) | 0 (0)
Blepharochalasis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 13 (13) | 11 (11)
Cataract Diabetic (Eye disorders) | 1 (1) | 0 (0)
Cataract Subcapsular (Eye disorders) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Corneal Degeneration (Eye disorders) | 1 (1) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Eye Muscle Entrapment (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 2 (2)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)
Ocular Myasthenia (Eye disorders) | 1 (1) | 0 (0)
Optic Ischaemic Neuropathy (Eye disorders) | 1 (1) | 1 (1)
Posterior Capsule Opacification (Eye disorders) | 1 (1) | 0 (0)
Retinal Artery Embolism (Eye disorders) | 1 (1) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 1 (1) | 2 (2)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 1 (1)
Ulcerative Keratitis (Eye disorders) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0)
Vitreous Detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Abdominal Adhesions (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 5 (5) | 4 (4)
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 12 (12) | 9 (10)
Abdominal Pain Upper (Gastrointestinal disorders) | 6 (6) | 9 (9)
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 2 (2) | 1 (1)
Alcoholic Pancreatitis (Gastrointestinal disorders) | 3 (4) | 5 (5)
Anal Fissure (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal Incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendix Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's Oesophagus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Bile Acid Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breath Odour (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Colitis (Gastrointestinal disorders) | 7 (7) | 2 (2)
Colitis Ischaemic (Gastrointestinal disorders) | 6 (6) | 1 (1)
Colitis Microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic Gastroparesis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (4)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dieulafoy's Vascular Malformation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 4 (4) | 6 (8)
Duodenal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 5 (5) | 3 (3)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 9 (10) | 4 (4)
Duodenal Vascular Ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenitis Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 4 (4)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral Hernia, Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fistula Of Small Intestine (Gastrointestinal disorders) | 0 (0) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Polyps (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric Ulcer (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 11 (12) | 14 (14)
Gastric Ulcer, Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 17 (19) | 11 (11)
Gastritis Erosive (Gastrointestinal disorders) | 3 (3) | 7 (7)
Gastritis Haemorrhagic (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis Haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Angiectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 13 (13) | 11 (12)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Mucosal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Polyp Haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 19 (20) | 21 (24)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 5 (5)
Hiatus Hernia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Hiatus Hernia Strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 2 (2)
Ileus Paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Inguinal Hernia (Gastrointestinal disorders) | 15 (15) | 29 (29)
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (3) | 2 (2)
Intestinal Obstruction (Gastrointestinal disorders) | 6 (7) | 5 (5)
Intestinal Perforation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Large Intestine Polyp (Gastrointestinal disorders) | 2 (2) | 4 (4)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Lumbar Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 (1) | 3 (3)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric Panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Obstruction Gastric (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 2 (2) | 5 (7)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Rupture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Failure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 6 (6) | 3 (3)
Pancreatitis Acute (Gastrointestinal disorders) | 16 (16) | 15 (15)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 (1) | 3 (3)
Peptic Ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritoneal Cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 4 (6) | 2 (2)
Rectal Prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary Duct Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary Gland Calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 (6) | 7 (7)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small Intestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen Tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 7 (7) | 7 (7)
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 7 (8) | 6 (6)
Varices Oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 5 (5)
Asthenia (General disorders) | 3 (3) | 6 (6)
Chest Discomfort (General disorders) | 5 (5) | 4 (4)
Chest Pain (General disorders) | 29 (32) | 25 (27)
Death (General disorders) | 33 (33) | 25 (25)
Device Related Thrombosis (General disorders) | 0 (0) | 1 (1)
Exercise Tolerance Decreased (General disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 3 (4) | 1 (1)
Implant Site Haematoma (General disorders) | 1 (1) | 0 (0)
Implant Site Pain (General disorders) | 1 (1) | 1 (1)
Incarcerated Hernia (General disorders) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 2 (2)
Injection Site Reaction (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 1 (1)
Medical Device Pain (General disorders) | 1 (1) | 0 (0)
Medical Device Site Dermatitis (General disorders) | 1 (1) | 0 (0)
Medical Device Site Joint Pain (General disorders) | 1 (1) | 0 (0)
Medical Device Site Pain (General disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 8 (8) | 5 (5)
Non-Cardiac Chest Pain (General disorders) | 222 (256) | 219 (264)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2)
Pacemaker Generated Arrhythmia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pelvic Mass (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 6 (6)
Soft Tissue Inflammation (General disorders) | 0 (0) | 1 (1)
Strangulated Hernia (General disorders) | 1 (1) | 0 (0)
Sudden Cardiac Death (General disorders) | 42 (42) | 36 (36)
Sudden Death (General disorders) | 9 (9) | 14 (14)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0)
Vascular Stent Restenosis (General disorders) | 1 (1) | 9 (9)
Vascular Stent Thrombosis (General disorders) | 2 (2) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 2 (2) | 0 (0)
Vessel Puncture Site Haemorrhage (General disorders) | 1 (1) | 0 (0)
Acute Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ampulla Of Vater Stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile Duct Stenosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile Duct Stone (Hepatobiliary disorders) | 7 (7) | 3 (3)
Biliary Colic (Hepatobiliary disorders) | 3 (3) | 2 (2)
Biliary Dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary Tract Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholangitis Acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis Sclerosing (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 14 (14) | 8 (9)
Cholecystitis Acute (Hepatobiliary disorders) | 14 (14) | 11 (11)
Cholecystitis Chronic (Hepatobiliary disorders) | 6 (6) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 35 (35) | 25 (25)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Chronic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 6 (6) | 15 (15)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic Congestion (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic Vein Dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis Alcoholic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis Chronic Active (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis Toxic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperplastic Cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic Hepatitis (Hepatobiliary disorders) | 3 (3) | 3 (4)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Liver Disorder (Hepatobiliary disorders) | 1 (1) | 2 (2)
Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy To Arthropod Bite (Immune system disorders) | 1 (1) | 0 (0)
Allergy To Arthropod Sting (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 2 (2) | 4 (4)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 2 (2)
Contrast Media Allergy (Immune system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Iodine Allergy (Immune system disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 3 (3)
Abdominal Infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 4 (4) | 4 (4)
Acute Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Acute Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 4 (4)
Appendiceal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 10 (10) | 13 (13)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 2 (2)
Atypical Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial Prostatitis (Infections and infestations) | 2 (2) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bone Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Borrelia Infection (Infections and infestations) | 0 (0) | 1 (1)
Breast Abscess (Infections and infestations) | 1 (1) | 1 (1)
Breast Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 17 (21) | 16 (17)
Bronchitis Bacterial (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis Viral (Infections and infestations) | 1 (2) | 2 (2)
Brucellosis (Infections and infestations) | 0 (0) | 1 (1)
Bursitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Candida Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 37 (40) | 32 (35)
Cellulitis Of Male External Genital Organ (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis Staphylococcal (Infections and infestations) | 2 (2) | 1 (1)
Cholangitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis Infective (Infections and infestations) | 2 (2) | 7 (7)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Citrobacter Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 3 (3) | 3 (3)
Cutaneous Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 2 (2)
Cytomegalovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Dengue Fever (Infections and infestations) | 8 (8) | 3 (3)
Dermo-Hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 2 (2) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 5 (5) | 1 (1)
Diabetic Gangrene (Infections and infestations) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 10 (11) | 9 (9)
Diverticulitis Intestinal Haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Enterobacter Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis Infectious (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 8 (9) | 7 (7)
Escherichia Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Escherichia Urinary Tract Infection (Infections and infestations) | 3 (3) | 6 (6)
External Ear Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Extradural Abscess (Infections and infestations) | 0 (0) | 2 (2)
Gallbladder Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 6 (6) | 4 (4)
Gastric Ulcer Helicobacter (Infections and infestations) | 0 (0) | 1 (1)
Gastritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 25 (25) | 26 (31)
Gastroenteritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Salmonella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 3 (3) | 2 (2)
Graft Infection (Infections and infestations) | 1 (1) | 0 (0)
Groin Abscess (Infections and infestations) | 2 (2) | 2 (2)
Haemophilus Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hantaviral Infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter Gastritis (Infections and infestations) | 1 (1) | 1 (1)
Hepatic Amoebiasis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 1 (1)
Herpes Virus Infection (Infections and infestations) | 0 (0) | 2 (2)
Herpes Zoster (Infections and infestations) | 0 (0) | 4 (4)
Iatrogenic Infection (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Infected Bite (Infections and infestations) | 0 (0) | 1 (1)
Infected Cyst (Infections and infestations) | 2 (2) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious Colitis (Infections and infestations) | 4 (4) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 1 (1)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 7 (9) | 11 (12)
Influenza (Infections and infestations) | 5 (5) | 5 (5)
Injection Site Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Latent Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Liver Abscess (Infections and infestations) | 1 (1) | 1 (1)
Localised Infection (Infections and infestations) | 5 (5) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 10 (10) | 11 (12)
Ludwig Angina (Infections and infestations) | 0 (0) | 1 (1)
Lung Abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 5 (6)
Lyme Disease (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Medical Device Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Aseptic (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Necrotising Fasciitis (Infections and infestations) | 1 (1) | 3 (3)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 2 (2) | 2 (2)
Osteomyelitis (Infections and infestations) | 8 (13) | 5 (6)
Osteomyelitis Acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis Chronic (Infections and infestations) | 1 (1) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media Acute (Infections and infestations) | 0 (0) | 2 (2)
Pancreas Infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pelvic Inflammatory Disease (Infections and infestations) | 0 (0) | 1 (1)
Perichondritis (Infections and infestations) | 3 (3) | 0 (0)
Perihepatic Abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal Abscess (Infections and infestations) | 1 (2) | 1 (1)
Peritoneal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 5 (5)
Peritonsillar Abscess (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngolaryngeal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal Cyst (Infections and infestations) | 0 (0) | 2 (2)
Pleurisy Viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 108 (123) | 96 (98)
Pneumonia Bacterial (Infections and infestations) | 3 (3) | 5 (5)
Pneumonia Chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Klebsiella (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Legionella (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia Mycoplasmal (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia Pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Viral (Infections and infestations) | 3 (3) | 1 (1)
Post Procedural Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Post Procedural Infection (Infections and infestations) | 2 (2) | 2 (2)
Post Procedural Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post Procedural Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Post Viral Fatigue Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 13 (14) | 13 (13)
Proctitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous Colitis (Infections and infestations) | 2 (2) | 1 (1)
Pseudomonal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Psoas Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Pulmonary Tuberculosis (Infections and infestations) | 4 (4) | 3 (3)
Pyelonephritis (Infections and infestations) | 9 (9) | 4 (4)
Pyelonephritis Acute (Infections and infestations) | 5 (5) | 6 (6)
Pyelonephritis Chronic (Infections and infestations) | 1 (1) | 1 (2)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 4 (4) | 1 (1)
Scrotal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Scrub Typhus (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 35 (38) | 20 (20)
Septic Shock (Infections and infestations) | 12 (13) | 11 (11)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 5 (5) | 6 (6)
Systemic Infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 5 (5) | 0 (0)
Toxic Shock Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculous Pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (9) | 7 (7)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 33 (35) | 27 (28)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection Staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 10 (11) | 16 (16)
Vestibular Neuronitis (Infections and infestations) | 3 (3) | 2 (2)
Viral Cardiomyopathy (Infections and infestations) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 6 (6) | 8 (8)
Viral Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Myocarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral Pericarditis (Infections and infestations) | 1 (1) | 3 (3)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (3)
Visceral Leishmaniasis (Infections and infestations) | 1 (1) | 0 (0)
Vulval Abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 4 (4) | 0 (0)
Wound Infection Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 9 (14) | 8 (8)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Anaesthetic Complication Neurological (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 8 (9) | 7 (7)
Aortic Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial Bypass Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod Sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Auricular Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blast Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brachial Plexus Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Brain Herniation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cardiac Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac Valve Replacement Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Chemical Burn Of Gastrointestinal Tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 8 (8) | 2 (2)
Confusion Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (6) | 3 (3)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Delayed Recovery From Anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electric Shock (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Extra-Axial Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 32 (34) | 26 (26)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Femur Fracture (Injury, poisoning and procedural complications) | 9 (9) | 13 (14)
Fibula Fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foreign Body In Urogenital Tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture Displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured Skull Depressed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Stoma Necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Heat Stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2) | 7 (8)
Humerus Fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 8 (18) | 6 (6)
Jaw Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Mallet Finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 3 (5) | 6 (7)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Multiple Injuries (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Muscle Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Rupture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Nerve Root Injury Lumbar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oesophageal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Penetrating Abdominal Trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirenal Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Post Concussion Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Fistula (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 8 (8) | 7 (7)
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Pulmonary Embolism (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post Procedural Swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Pubis Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Radiation Associated Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation Skin Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Rib Fracture (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Road Traffic Accident (Injury, poisoning and procedural complications) | 19 (19) | 14 (14)
Scapula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Silicosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Skin Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Spinal Cord Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Splenic Rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma Site Discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomal Hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Tendon Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Tracheostomy Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Traumatic Haemothorax (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Renal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Access Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Vascular Pseudoaneurysm Ruptured (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 11 (11) | 10 (10)
Anticoagulation Drug Level Above Therapeutic (Investigations) | 2 (2) | 0 (0)
Blood Calcium Increased (Investigations) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Mb Increased (Investigations) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 4 (4) | 5 (5)
Blood Creatinine Increased (Investigations) | 2 (2) | 0 (0)
Blood Potassium Increased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Brain Natriuretic Peptide Increased (Investigations) | 0 (0) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Cardiac Stress Test Abnormal (Investigations) | 1 (1) | 0 (0)
Ejection Fraction Decreased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0)
Exercise Electrocardiogram Abnormal (Investigations) | 1 (1) | 1 (1)
Glomerular Filtration Rate Decreased (Investigations) | 1 (1) | 0 (0)
Hiv Test Positive (Investigations) | 1 (1) | 0 (0)
Haematocrit Decreased (Investigations) | 0 (0) | 1 (1)
Haematocrit Increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 1 (1) | 1 (1)
Hepatic Enzyme Abnormal (Investigations) | 0 (0) | 2 (2)
Hepatic Enzyme Increased (Investigations) | 3 (3) | 5 (5)
Hepatitis C Virus Test Positive (Investigations) | 0 (0) | 1 (1)
Human Papilloma Virus Test Positive (Investigations) | 0 (0) | 1 (1)
Influenza A Virus Test Positive (Investigations) | 0 (0) | 1 (1)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 3 (3) | 1 (1)
Liver Function Test Increased (Investigations) | 3 (3) | 1 (1)
Mycobacterium Tuberculosis Complex Test Positive (Investigations) | 2 (2) | 0 (0)
Scan Myocardial Perfusion (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 3 (3) | 5 (5)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Tumour Marker Increased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 2 (2) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 13 (13) | 13 (14)
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 16 (21) | 20 (20)
Diabetic Complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 9 (13) | 4 (4)
Diabetic Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Fluid Overload (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Fluid Retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (9) | 10 (12)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperinsulinaemic Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (12) | 8 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Metabolic Disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 36 (36) | 37 (37)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 9 (10)
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femoroacetabular Impingement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 21 (22) | 21 (21)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10)
Meniscal Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 35 (44) | 24 (26)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 46 (51) | 50 (54)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Rheumatic Fever (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (10)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal Ligament Ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Sympathetic Posterior Cervical Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 10 (10)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaplastic Large Cell Lymphoma T- And Null-Cell Types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-Cell Small Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (18) | 11 (12)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bladder Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 8 (8)
Bladder Transitional Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Breast Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carcinoid Tumour Of The Appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cardiac Myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac Valve Fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Colon Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ductal Adenocarcinoma Of Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrooesophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma Of Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hair Follicle Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's Disease Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Inflammatory Pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 8 (8)
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Large Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Lung Adenocarcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung Adenocarcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung Adenocarcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung Adenocarcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Lung Squamous Cell Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung Squamous Cell Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung Squamous Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung Squamous Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung Squamous Cell Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant Anorectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Malignant Melanoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant Melanoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Palate Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Sweat Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Metastases To Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Carcinoma Of The Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Monoclonal Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mucinous Cystadenocarcinoma Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine Tumour Of The Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine Tumour Of The Lung Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Non-Hodgkin's Lymphoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Small Cell Lung Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Small Cell Lung Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Oesophageal Adenocarcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatic Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penile Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peritoneal Mesothelioma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17) | 18 (18)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Prostate Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
Prostate Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Prostate Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Prostate Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectal Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cell Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Salivary Gland Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sinonasal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sinus Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small Cell Lung Cancer Limited Stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 2 (2)
Squamous Cell Carcinoma Of The Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous Cell Carcinoma Of The Hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of The Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous Cell Carcinoma Of The Vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Synovial Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Transitional Cell Cancer Of Renal Pelvis And Ureter Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Urinary Bladder Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Vocal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alcoholic Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 3 (3) | 4 (4)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic Nervous System Imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Axonal Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Balance Disorder (Nervous system disorders) | 1 (1) | 2 (2)
Brain Injury (Nervous system disorders) | 0 (0) | 2 (2)
Brain Oedema (Nervous system disorders) | 1 (1) | 1 (1)
Carotid Arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Disease (Nervous system disorders) | 1 (1) | 1 (1)
Carotid Artery Occlusion (Nervous system disorders) | 3 (3) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 19 (19) | 14 (14)
Carotid Artery Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Sinus Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 6 (6) | 6 (6)
Cauda Equina Syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral Atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrospinal Fistula (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1)
Cervical Radiculopathy (Nervous system disorders) | 2 (2) | 2 (2)
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 2 (2) | 3 (3)
Coordination Abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Cubital Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 4 (4)
Dementia Alzheimer's Type (Nervous system disorders) | 1 (1) | 1 (1)
Demyelinating Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic Neuropathy (Nervous system disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 8 (8) | 7 (7)
Dizziness Exertional (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 3 (3) | 5 (7)
Epilepsy (Nervous system disorders) | 6 (7) | 5 (5)
Epileptic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Essential Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial Paralysis (Nervous system disorders) | 2 (2) | 2 (2)
Focal Dyscognitive Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 2 (3) | 2 (2)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 4 (4)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (3) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycaemic Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 2 (2)
Hypoglycaemic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatraemic Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 4 (4) | 1 (1)
Intercostal Neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial Mass (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Venous Sinus Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 2 (2)
Limbic Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 8 (8) | 6 (8)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Lumbosacral Radiculopathy (Nervous system disorders) | 2 (2) | 2 (2)
Memory Impairment (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 2 (2) | 7 (7)
Migraine (Nervous system disorders) | 3 (3) | 1 (1)
Migraine With Aura (Nervous system disorders) | 1 (1) | 0 (0)
Mixed Dementia (Nervous system disorders) | 0 (0) | 2 (2)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 2 (3) | 1 (2)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Nerve Compression (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuromuscular Pain (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 4 (4) | 0 (0)
Occipital Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 8 (8) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 4 (4)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures With Secondary Generalisation (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral Nerve Lesion (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Petit Mal Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Postictal Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 9 (9)
Pyramidal Tract Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radial Nerve Palsy (Nervous system disorders) | 0 (0) | 2 (2)
Radicular Pain (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 2 (3)
Ruptured Cerebral Aneurysm (Nervous system disorders) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 6 (6)
Seizure (Nervous system disorders) | 7 (7) | 5 (5)
Sensory Loss (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 2 (2) | 0 (0)
Spondylitic Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 73 (82) | 67 (73)
Toxic Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Transient Global Amnesia (Nervous system disorders) | 0 (0) | 3 (3)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ulnar Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Ulnar Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Vith Nerve Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vith Nerve Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Vascular Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral Artery Occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar Insufficiency (Nervous system disorders) | 2 (2) | 0 (0)
Vertigo Cns Origin (Nervous system disorders) | 1 (1) | 0 (0)
Device Dislocation (Product Issues) | 1 (3) | 2 (2)
Device Lead Damage (Product Issues) | 0 (0) | 1 (1)
Device Malfunction (Product Issues) | 1 (1) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 1 (1)
Lead Dislodgement (Product Issues) | 0 (0) | 1 (1)
Thrombosis In Device (Product Issues) | 0 (0) | 1 (2)
Acute Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment Disorder With Mixed Disturbance Of Emotion And Conduct (Psychiatric disorders) | 1 (1) | 0 (0)
Affective Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Agoraphobia (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 2 (2) | 6 (6)
Alcoholic Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 1 (1)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (9) | 3 (3)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Borderline Personality Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bradyphrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 6 (6) | 3 (3)
Confusional State (Psychiatric disorders) | 3 (3) | 1 (1)
Conversion Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 3 (3)
Delirium Tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Delusional Disorder, Unspecified Type (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 25 (26) | 13 (18)
Depression Suicidal (Psychiatric disorders) | 3 (3) | 0 (0)
Drug Abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Factitious Disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal Ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Major Depression (Psychiatric disorders) | 2 (2) | 5 (5)
Mental Status Changes (Psychiatric disorders) | 4 (4) | 7 (10)
Mood Disorder Due To A General Medical Condition (Psychiatric disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 1 (1)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 8 (10) | 7 (7)
Suicide Attempt (Psychiatric disorders) | 14 (15) | 5 (5)
Transient Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 62 (74) | 57 (59)
Acute Prerenal Failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Bladder Dilatation (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Outlet Obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Bladder Perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder Tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 2 (2)
Chronic Kidney Disease (Renal and urinary disorders) | 15 (16) | 13 (14)
Cystitis Glandularis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis Interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis Noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic Cystopathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 3 (3)
End Stage Renal Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis Proliferative (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 13 (15) | 9 (9)
Hydronephrosis (Renal and urinary disorders) | 6 (7) | 2 (2)
Hypertensive Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Iga Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 21 (21) | 15 (15)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy Toxic (Renal and urinary disorders) | 6 (6) | 10 (10)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 2 (2)
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Postrenal Failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal Artery Occlusion (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Artery Stenosis (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal Colic (Renal and urinary disorders) | 6 (6) | 4 (4)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Cyst Haemorrhage (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 6 (6) | 8 (8)
Renal Haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 2 (4) | 0 (0)
Renal Infarct (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Tubular Disorder (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Vein Thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteral Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric Stenosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 15 (15) | 12 (14)
Urethral Stenosis (Renal and urinary disorders) | 0 (0) | 4 (5)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Bladder Rupture (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 3 (3) | 3 (3)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital Fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired Hydrocele (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Acquired Phimosis (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 13 (13) | 16 (16)
Breast Mass (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Peyronie's Disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal Ulcer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterovaginal Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vulva Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acquired Diaphragmatic Eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 24 (35) | 19 (21)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 10 (10)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 51 (76) | 38 (47)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 20 (21)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 10 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Laryngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal Mucosal Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal Turbinate Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (9)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Calcification (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 16 (16)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 8 (11)
Respiratory Tract Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal Cord Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 7 (8) | 4 (4)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 11 (11) | 6 (6)
Diabetic Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Reaction With Eosinophilia And Systemic Symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema Nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scar Pain (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Urticaria Chronic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vascular Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Physical Assault (Social circumstances) | 0 (0) | 1 (1)
Accelerated Hypertension (Vascular disorders) | 4 (4) | 3 (3)
Aortic Aneurysm (Vascular disorders) | 12 (12) | 10 (10)
Aortic Aneurysm Rupture (Vascular disorders) | 2 (2) | 1 (1)
Aortic Dissection (Vascular disorders) | 2 (2) | 1 (1)
Aortic Intramural Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Aorto-Duodenal Fistula (Vascular disorders) | 1 (1) | 1 (1)
Arterial Insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 3 (3)
Blood Pressure Inadequately Controlled (Vascular disorders) | 0 (0) | 1 (1)
Circulatory Collapse (Vascular disorders) | 2 (2) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 8 (9) | 11 (13)
Dry Gangrene (Vascular disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Embolism Venous (Vascular disorders) | 1 (1) | 0 (0)
Essential Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Extremity Necrosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 3 (3)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 36 (41) | 34 (35)
Hypertensive Crisis (Vascular disorders) | 17 (19) | 21 (22)
Hypertensive Emergency (Vascular disorders) | 4 (7) | 3 (3)
Hypotension (Vascular disorders) | 17 (17) | 16 (16)
Hypovolaemic Shock (Vascular disorders) | 3 (3) | 1 (1)
Iliac Artery Embolism (Vascular disorders) | 0 (0) | 1 (1)
Iliac Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Intermittent Claudication (Vascular disorders) | 6 (7) | 4 (4)
Ischaemic Limb Pain (Vascular disorders) | 0 (0) | 2 (2)
Leriche Syndrome (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic Fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
Malignant Hypertension (Vascular disorders) | 3 (4) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Penetrating Aortic Ulcer (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 47 (49) | 27 (29)
Peripheral Artery Aneurysm (Vascular disorders) | 2 (2) | 5 (6)
Peripheral Artery Dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Occlusion (Vascular disorders) | 13 (15) | 7 (7)
Peripheral Artery Stenosis (Vascular disorders) | 8 (11) | 8 (9)
Peripheral Artery Thrombosis (Vascular disorders) | 4 (5) | 1 (1)
Peripheral Embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 20 (23) | 7 (7)
Peripheral Vascular Disorder (Vascular disorders) | 6 (6) | 3 (3)
Peripheral Venous Disease (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's Phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Renovascular Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 3 (3)
Shock Haemorrhagic (Vascular disorders) | 4 (4) | 1 (1)
Subclavian Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Subclavian Artery Stenosis (Vascular disorders) | 2 (2) | 1 (1)
Superior Vena Cava Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Temporal Arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 3 (3) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose Vein (Vascular disorders) | 3 (3) | 0 (0)
Venous Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9443) | Alirocumab (N=9451)
Non-Cardiac Chest Pain (General disorders) | 462 (556) | 481 (591)
Nasopharyngitis (Infections and infestations) | 532 (697) | 567 (713)
Blood Creatine Phosphokinase Increased (Investigations) | 488 (560) | 457 (521)
Myalgia (Musculoskeletal and connective tissue disorders) | 496 (563) | 522 (591)
Hypertension (Vascular disorders) | 574 (678) | 542 (600)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT01663402/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT01663402/SAP_001.pdf